## TWILIGHT Study: Treatment with Light Therapy

Effect of light exposure during acute rehabilitation on sleep after traumatic brain injury

Protocol Version 1.2

Funded by National Institute on Disability and Rehabilitation Research (NIDRR)

H133A120028 H133G120055 H133A120084

## **Confidentiality Statement**

This document is confidential and is to be distributed for review only to investigators, potential investigators, consultants, study staff, and applicable independent ethics committees or institutional review boards. The contents of this document shall not be disclosed to others without written authorization unless it is necessary to obtain informed consent from potential study participants.

## University of Washington TBI Model System (TBIMS) Group:

| Jeanne M. Hoffman, Ph.D. | Principal Investigator | jeanneh@uw.edu |
|--------------------------------|---------------------------|-----------------|
| Donald Fogelberg, Ph.D., OTR/L | Investigator | fogelber@uw.edu |
| Jennifer Zumsteg, M.D. | Investigator | zumsteg@uw.edu |
| Sureyya Dikmen, Ph.D. | Investigator | dikmen@uw.edu |
| Rena Reyes, M.D. | Data Safety Monitor | rreyes@uw.edu |
| Jason Barber, M.S. | Data Analyst/Statistician | barber@uw.edu |
| Erica Wasmund | Research Coordinator | ericaw8@uw.edu |

#### **University of Texas Southwestern**

Kathleen R. Bell, M.D. Investigator Kathleen.Bell@UTSouthwestern.edu

## Mount Sinai, New York TBIMS Group:

Jason Krellman Principal Investigator

Anne F. Ambrose, M.D. Investigator

Tausif Billah, B.A. Research Coordinator Michelle Urman Research Coordinator

### **Baylor Institute for Rehabilitation, North Texas TBIMS Group:**

Randi Dubiel, D.O. Principal Investigator

Shahid Shafi, M.D., MPH Investigator

Cindy Dunklin, B.S., CCRC Project Coordinator

## James A. Haley Veterans Hospital

Risa Nakase-Richardson, Ph.D. Study Consultant/Investigator

#### **Project Officer, NIDRR:**

Cate Miller, Ph.D. Cate.Miller@ed.gov

| TABLE OF CONTENTS | Page |
|---|---|
| Title/Investigators | 1 |
| Table of Contents | 2 |
| Background and Significance | 3-4 |
| Target Population | 4 |
| Potential benefit to this population | 4 |
| Research Hypotheses and Specific Aims | 4<br>5 |
| Study Description | 5-6 |
| Figure 1: Summary Overview of Study Procedures for TWILIGHT | 6 |
| Screening/Study Sample | 6 |
| Inclusion Criteria | 7 |
| Exclusion Criteria | 7 |
| Rationale for Study Population | 7 |
| Data Collection and Measures | 7-10 |
| Table 1: Data Collection Measures and Areas Assessed | 8 |
| Study Procedures | 10-12 |
| Data Analysis | 12 |
| Data Management | 13-14 |
| Table 2: Performance Measures | |
| Safety and Adverse Events | 14 |
| Definitions | 14-15 |
| Recording of Adverse Events | 16 |
| Ethical Considerations/Protection of Human Subjects | 17-18 |
| Potential Risks, Potential Benefits, Intent to Benefit, and Risk/Benefit Ratio | 18-19 |
| Importance of Knowledge to be Gained | 19 |
| Overall Project Evaluation | 20 |
| List of Acronyms and Abbreviations | 21 |
| References and Works Cited | 22-30 |
| Appendix | 31-44 |

#### I. Background and Significance:

Sleep disturbance is a common clinical problem after Traumatic Brain Injury (TBI). Disrupted sleep exacerbates other symptoms after TBI such as fatigue and can impede overall recovery after TBI (Castriotta RJ W. M., June 15, 2007) (Mathias JL, 2012;13). Trouble falling or staying asleep (insomnia) and reversal of sleep/wake cycles (circadian rhythm disorders) are two categories of sleep disturbance occurring frequently after TBI. Insomnia affects roughly one-third of TBI survivors and reports of overall sleep disturbances are as high as 70% (Mathias JL, 2012;13). In a study by Ayalon et al. (Ayalon L, 2007), 36% of individuals with TBI who reported suffering from insomnia met the diagnostic criteria for a circadian rhythm sleep disorder. Sleep disturbances are also common during inpatient rehabilitation. Makley et al. (Makley MJ E. J., 2008) found that 68% of patients with a closed head injury demonstrated disturbed sleep during inpatient rehabilitation. The clinical utility of diagnosing sleep disorders using criteria from the Diagnostic and Statistical Manual or International Classification of Sleep Disorders is limited in clinical situations such as the first weeks of recovery after TBI as these diagnostic criteria require the presence of symptoms for at least a month, rely heavily on subjective report and can be confusing given the frequency of co-occurring medical and psychiatric disorders (Ohayon MM, 2009). In these clinical situations, other tools for assessing sleep quality may be especially useful. These tools include sleep logs, measurements of movement with actigraphy and overall clinical assessment of sleep patterns.

Most studies looking at treatment of sleep disturbances and wakefulness after TBI have focused on pharmacologic interventions and have reported limited efficacy in improving sleep. The sedative-hypnotic medications typically used in the treatment of sleep disorders in the general population are often not appropriate for use after TBI given concerns about cognitive and behavioral side effects (Flanagan SR, 2007) (Larson EB, 2010). There are case reports of improved sleep in the chronic phase of TBI recovery with cognitive behavioral therapy (Ouellet MC M. C., 2007) and light exposure (Carter KA, 2010) (Chesson AL, 1999) but these treatments have not been studied in the acute rehabilitation phase. BWL exposure is considered an appropriate option for some sleep disorders in a variety of clinical populations including those with dementia (Mishima K, 1994) (Riemersma-van der Lek RF, 2008). The proposed study will help elucidate both the effects of BWL exposure after TBI in the inpatient rehabilitation setting as well as clinical feasibility of delivering light exposure in this case setting.

Sleep disturbance may hinder the rehabilitation process. Clinically significant sleep disturbances after TBI correlate with higher rates of depression, anxiety, pain (Fogelberg DJ, 2012) and fatigue (Englander J, 2010), all conditions which could deter full engagement in rehabilitation. Even in a healthy population a moderate reduction in the amount of quality sleep over time can negatively impact cognitive functions such as behavioral alertness and working memory (Banks S, 2007). BWL exposure has been shown to be effective in both reducing agitated behavior and improving cognition in older adults with dementia (Mishima K, 1994) (Riemersma-van der Lek RF, 2008) (Forbes D, 2011). After TBI, there is an association of sleep problems with more functional limitations, higher reliance on other people for care, and diminished satisfaction with quality of life at one year after injury (Fogelberg DJ, 2012). Improved sleep in the acute recovery phase after TBI may positively impact other rehabilitation outcomes. In the study by Makley, et al. (Makley MJ J.-G. L., 2009) sleep disturbance was associated with longer average length of stay for both acute trauma center (22 days vs. 9 days) and inpatient rehabilitation (37 days vs. 21 days). In non-TBI populations BWL exposure has shown efficacy in the treatment of mood symptoms and improving alertness even with small doses and durations of treatment. such as a single one-hour session (Reeves GM, 2012) (Riemersma-van der Lek RF, 2008) (Revell VL, Jan 2006) (Chang AM, 2012) (Terman M, 2005) (Wirz-Justice A, 2012) (Friedman L, May 2012)

(Neikrug AB, 2012). These additional effects of BWL exposure may provide clinical benefit beyond improved sleep in persons recovering from TBI and will be assessed in the proposed study.

Research and clinical evaluation of sleep often employ actigraphy, which allows for the evaluation of subject movement over time and can be extrapolated to wake/rest cycles (Morgenthaler TI, 2007). Use of actigraphy for sleep evaluation with subjects after brain injury has been successful in both inpatient (Zollman FS C. C., 2010) and outpatient settings (Ayalon L, 2007). Additionally, considerations regarding movements and sleep specific to TBI and actigraph placement, including spasticity and paresis (Zollman FS C. C., 2010), are important and will be considered in the execution of this study.

Our study group has extensive experience with the inpatient Rehabilitation brain injured population, research experience in regards to sleep after brain injury, and demonstrated use of light therapy and actigraphy in individuals with TBI (Fogelberg DJ, 2012) (Watson NF, 2007). The University of Washington investigators have current IRB permission to conduct a pilot study of BWL exposure on the acute rehabilitation unit to allow for the current study protocol to be refined early in the research process and demonstrate logistics and feasibility to collaborating TBIMS centers. In the current health care climate, low cost treatments with low staff burden are valued and we will evaluate these factors in this study (Wood RL, 1999) (Whitmore RG, 2012).

## II. Target Population:

Individuals aged 18-70 years with moderate to severe traumatic brain injury (TBI), 30 days or less out from TBI hospitalized on acute inpatient rehabilitation. Moderate to severe TBI will be determined using the TBI Model System (TBIMS) case definition (Traumatic Brain Injury Model Systems, 2013): damage to brain tissue caused by an external mechanical force, post-traumatic amnesia (PTA) greater than 24 hours, or loss of consciousness greater than 30 minutes or Glasgow Coma Scale (GCS) score in the Emergency Department of 3-12, or intracranial abnormalities on imaging (Cuthbert JP, 2012).

Exclusion parameters for age and time since injury are needed in this study since sleep patterns and light effects change with aging and the focus of this study is in the early recovery phase of TBI. Potential subjects will be excluded from the study if they have a past medical history of bipolar disorder (Terman M, 2005); retinal pathology, complete blindness, or light sensitivity; absence of eye opening; tetraplegia with less than antigravity strength in all myotomes caudal to C6 level given the limitations on measuring movements with; or confirmed or suspected diagnosis of obstructive sleep apnea (Zollman FS C. C., 2010). BWL exposure is unlikely to change the underlying pathology for obstructed sleep and therefore potential subjects with a known history of sleep apnea treated with continuous positive pressure device, a body mass index > 40 kg/m2 at eligibility assessment, or who are classified as being "high risk" for sleep apnea based on the Berlin questionnaire (Netzer NC, 1999) will be excluded from the study. The Berlin questionnaire evaluates risks factors for sleep apnea including snoring, breathing pauses and daytime sleepiness. We are utilizing multiple criteria for exclusion for obstructive sleep apnea given the potential limitations of subjective questionnaires in subjects with TBI.

#### III. Potential benefit to this population:

Bright White Light (BWL) exposure has potential to clinically impact care for persons with Traumatic Brain Injury, especially given the prevalence of co-occurring conditions such as sleep and mood disorders. Investigations into the use and tolerance of Bright White Light exposure in this population are limited, especially in the acute recovery phase and in the inpatient setting. This study will improve our understanding of therapeutic and functional effects of light therapy and the relationship

with sleep efficiency. There is interest in non-pharmacologic treatment options for complications arising from patients experiencing a Traumatic Brain Injury (TBI), and this study investigates a treatment option and feasibility of integrating into usual care in the inpatient rehabilitation unit setting. If our hypothesis is correct, and there is clinically significant benefit from Bright White Light exposure, some study participants may have direct benefit from this study.

## IV. Research Hypothesis's and Specific Aims

## Specific Aims:

<u>Aim 1</u>: In persons with TBI, prospectively compare overnight sleep efficiency in a cohort exposed to morning Bright White Light with a comparison group exposed to Red Light in an acute inpatient rehabilitation setting.

<u>Aim 2</u>: Explore the relationship between Bright White Light exposure during inpatient rehabilitation after TBI and mood, therapy participation, attention, rate of functional recovery and length of stay.

<u>Aim 3</u>: Develop and describe sleep study procedures on the inpatient rehabilitation unit for persons with TBI to support optimal and feasible design of future studies in this important area.

## Research Hypothesis:

In persons with TBI, prospectively compare overnight sleep in a cohort exposed to morning Bright White Light with a comparison group exposed to Red Light in an acute inpatient rehabilitation setting.

<u>Hypothesis 1:</u> Individuals exposed to Bright White Light for 30 minutes each morning will have better sleep compared to the Red Light exposure group, as measured by sleep efficiency.

<u>Hypothesis 2:</u> Individuals with daily morning Bright White Light exposure will have better mood (as measured by the Positive and Negative Affective Schedule, PANAS), therapy participation (as measured by a 0-100 therapist rating) and attention (as measured by the Symbol Digit Modalities Test) at 10 days compared to individuals with daily Red Light exposure. The group exposed to Bright White Light will also have less daytime sleepiness and fatigue (as measured by the Karolinska Sleepiness Scale (KSS) and the Barrow Neurological Institute Fatigue Scale (BNI-FS), a faster rate of functional recovery as measured by FIM<sup>TM</sup> efficiency for the rehabilitation stay and a shorter length of stay compared to those in the Red Light group

<u>Hypothesis 3a:</u> Bright White Light exposure will be rated as a reasonable addition to clinical care by staff using Likert scale ratings. Categorize and quantify rates of any side effects of Bright White Light and Red Light exposure in persons with TBI during inpatient rehabilitation.

<u>Hypothesis 3b</u>: Bright White Light and Red Light exposure will be generally well tolerated with side effect profiles and rates similar to those observed in previous studies with other populations.

See Appendix for Flowchart on Specific Aims of this study

## V. Study Description

We propose to recruit a prospective cohort of persons with TBI to compare effects of Bright White Light exposure to Red Light (RL) exposure. Light therapy treatments will be given daily in the morning for up to 10 days, and an Actiwatch will be worn that records movements for the entirety of the study. We will utilize objective assessments of sleep quality, subjective mood report, rate sleepiness and fatigue and complete measures of attention and participation in rehabilitation therapies to explore the

effects of light exposure in the acute inpatient rehabilitation setting. We will also evaluate the anticipated device costs and staff burden involved in utilizing light therapy exposure in the inpatient rehabilitation clinical setting. An overview of study procedures with timeline is described in Figure 1 below with further details in the sections that follow.

Figure 1. Overview of Study Procedures for TWILIGHT



## VI. Screening for Eligibility:

Although subjects will be screened for this study concurrent with screening for eligibility for enrollment into the Traumatic Brain Injury Model System (TBIMS) study (Traumatic Brain Injury Model Systems, 2013), these are independent studies and subjects will have the choice to enroll in both, neither, or either one. The TBI Model Systems program, sponsored by the National Institute on Disability and Rehabilitation Research (NIDRR), is the largest longitudinal study of TBI in the nation. NIDRR awards 5 year grant awards to institutions that are national leaders in medical research and patient care and these. Institutions which receive this distinction are collectively termed, the TBI Model Systems. As part of the TBI Model Systems, the University of Washington TBI Model Systems research team is recognized as providing the highest level of comprehensive specialty services from the point of injury through chronic care stages, including re-entry into full community life. The current grant cycle is for the 2012-2017 time period, and one of the areas of interest for the UW TBI Model Systems research team is the treatment of sleep difficulties after TBI.

The screening process will begin will reviewing the medical charts for patients that are on the inpatient rehabilitation unit at Harborview Medical Center. If a patient meets the inclusion criteria, research staff will approach the patient to determine whether the patient is cognitively capable of giving their consent for the study by administering the Galveston Orientation and Amnesia Test. The study will then be explained to the patient; or if the patient is experiencing post traumatic amnesia, the study will be explained to the patient's legally authorized representative. Consent will be obtained either from the patient or, if he or she is unable to provide informed consent, the patient's legally authorized representative.

## VII. Study Sample:

Study participants will be recruited from acute inpatient rehabilitation at three participating TBI Model Systems institutions (University of Washington, Mount Sinai, Baylor). Eligible participants will be within three months of sustaining a moderate to severe TBI (as defined by the TBI Model Systems (Traumatic Brain Injury Model Systems, 2013)), admitted to acute inpatient rehabilitation, English speaking, and aged 18-70 years. Exclusionary medical factors will be identified in the medical record and through interview during screening/baseline assessment. In a pilot study comparing the effects of BWL and RL exposure in a sample of subjects with chronic TBI, Cantor et al. (Cantor, et al., 2012) reported an effect size of 0.63 for sleep duration. Because this pilot study involved subjects in the chronic phase of TBI, who were living at home rather than in an institution, and underwent a longer course of treatment (28 days in that study vs. 10 days in this study), we chose to take a conservative approach to calculating the required sample size. Based on an estimated effect size of 0.5 and 80% power, 128 subjects would be required to complete this study (64 per group). We anticipate recruitment over three years at three sites. Historical TBIMS and associated trial enrollment totals from the participating sites supports this study enrollment goal.

#### VIII. Inclusion Criteria:

- 1. Within three months of moderate to severe TBI
- 2. Admitted to acute inpatient rehabilitation
- 3. Ages 18-70
- 4. English speaking

#### VIII. Exclusion Criteria:

- 1. Complete blindness
- 2. Absence of eye opening or disorders of consciousness (Rancho level of 1-3)
- 3. Past medical history of retinal pathology
- 4. Past medical history of light sensitivity
- 5. Past medical history of narcolepsy
- 6. Past medical history of bipolar disorder
- 7. Past medical history of obstructive sleep apnea (OSA)
- 8. Sleep disturbance defined as having a "0" rating by research staff (using all sources available). If rated a "0" for no sleep disturbance, they must also NOT be receiving sleep medications in the last 72 hours
- 9. Suspected diagnosis of obstructive sleep apnea (determined by the Berlin Questionnaire)
- 10. Tetraplegia with less than antigravity strength in all myotomes caudal to C6 level given the limitations on measuring movements with actigraphy in this population (i.e. cannot reliably detect upper extremity or lower extremity movement with this level of paralysis).
- 11. Current medical orders indicated for night time sleep disruption (e.g. chest PT, MIE q2 hours of meds that disrupt sleep). \*May be re-approached if the medical orders are no longer in place.

#### IX. Rationale for Study Population

The study population of interest is TBI in the setting of acute inpatient rehabilitation, which is typically moderate to severe TBI. Persons less than 18 years of age or greater than 70 years are being excluded from the study because of baseline sleep physiology differences seen in younger and advanced ages. We wish to enroll those with sleep disturbances; those with normal sleep will not be enrolled. We are excluding those who would not benefit from light exposure due to eye abnormalities or those with other pathology that will interfere with sleep and cannot be affected by light exposure. Additionally, since actigraphy relies on limb movement for recording, those with tetraplegia would be excluded.

#### X. Data Collection and Measures

Screening of subjects will need to occur to determine eligibility of subjects, including review of medical chart. If patients are not eligible or are excluded based on exclusion criteria, no identifiable data is retained. Once consented into the study, the exclusion criteria will be reviewed with the patient and/or their legal representative. Data collection measures, areas assessed, and the timing of when this data is collected is shown in Table 1.

**Table 1: Data Collection Measures and Areas Assessed** 

| Measure | Area to be Assessed | Screening and | Intervention | Outcome |
|---|---|---|---|---|
| | | Baseline | | |
| | | (Day 0-2) | (Days 3-12) | (Day 13) |
| Demographics | Characteristics (age, | X | | |
| | education, gender) | | | |
| Injury characteristics | Cause of injury, date of | X | | |
| | injury, lowest GCS, | | | |
| | PTA/GOAT | | | |
| Medical History | Diagnoses, medications | X | | |
| | at enrollment, symptoms, | | | |
| | associated injuries (ICD- | | | |
| Berlin questionnaire | 9 codes), vital signs Sleep apnea | X | | |
| Clinician Rating: | Sleep disturbance | X | | |
| Delirium Rating Scale | Sleep disturbance | A | | |
| Revised 98 Item 1 | | | | |
| Makley scale | Sleep disturbance | X | X | |
| Actigraphy | Sleep parameters | X | X | |
| Light Therapy Time | Light exposure time | | X | |
| Medication categories | Potential confounders (see data sheet) | X | | X |
| FIM <sup>TM</sup> Scores and | Functional score | X | | X |
| Efficiency | | | | |
| Hospitalization | Acute LOS, Rehab LOS | X | | X |
| Symbol Digit | Attention | X | | X |
| Modalities Test | | | | |
| PANAS | Mood | X | | X |
| Therapy participation | Function | X | | X |
| Karolinska Sleepiness | Daytime sleepiness | X | | X |
| Scale | | | | |
| Barrow Neurological | Daytime fatigue | X | | X |
| Institute Fatigue Scale | | | | |

## A. Screening Measures:

The following data will be used as descriptive characteristics of the subjects upon study completion. Initially this data will be used during the screening process to ensure appropriate patients are approached for participation:

• **Demographics**: Age, gender, race/ethnicity, weight (kg), height (cm), BMI (calculated).

- **Injury Characteristics:** Time since injury, Post-resuscitation GCS score, duration of PTA as measured by TBIMS procedures using the Galveston Orientation and Amnesia Test (GOAT), associated injuries including ICD codes.
- **Medical History:** Current diagnoses, past diagnoses, medications (at enrollment, during treatment and at outcome measure), vital signs.
- **Berlin Questionnaire** (Netzer NC, 1999): The 10-item questionnaire consists of 3 categories related to the risk of having sleep apnea. Patients can be classified into High Risk or Low Risk based on their responses to the individual items and their overall scores in the symptom categories.

## **B.** Randomization Measure:

Randomization will occur by research staff member assessing the patient for sleep disturbance, using all sources available, in the first item question from the *Clinician Rating: Delirium Rating Scale – Revised 98* (DelRS-R98) (Trzepacz PT, 2001). Our recent prevalence work showed that 86% of acute TBI admissions have sleep abnormalities using clinician ratings, specifically the DelRS-R98 (Nakase-Richardson R S. M., Prospective evaluation of the nature, course, and impact of acute sleep abnormality following TBI, 2013). Sleep disturbance questions will be asked of the clinical staff whom were involved in caring for the patient during Day 1 of study participation, significant other (if available), and directly of the patient (if possible). The rating will be used as a sleep disturbance severity marker which will be utilized by the statistician during randomization to help control for sleep disturbance severity (Sjösten N, July 2009).

## C. Primary Outcome Measure:

Sleep efficiency scores derived from actigraphy data will be the primary outcome, and analysis will be done by Donald Fogelberg, Ph.D at the University of Washington. An Actiwatch 2 (Philips/Respironics, Bend, OR) will be used for study purposes to facilitate consistent measurement across sites. We will set the Actiwatch to record activity data in 60-second intervals. Actigraphy data will be automatically scored with Actiware software (Respironics, Philips Healthcare), which uses validated algorithms to determine whether an epoch of activity is "sleep" or "wake" (Cole RJ, 1992). Typically there is a lack of a consistent sleep/wake cycle in the study population, therefore we will be using sleep efficiency and total sleep time scores obtained during a set night-time interval (2200 to 0600) as the primary index of sleep function, as has been used in previous publications[39, 40]. We will be comparing average between group differences between the BWL and RL groups at baseline and after 10 days of light exposure.

#### **D. Secondary Outcome Measures:**

- Makley Scale: The Makley scale is a 4-point ordinal scale which allows staff to score sleep as follows: 0 = asleep; 1 = drowsy/falling asleep; 2 = drowsy/waking up; 3 = awake. An hourly sleep log on each patient will be filled out every two hours by the unit nursing staff from 2200 to 0600 hours starting at baseline and through the duration of the study.[41]]
- [42] Functional Independence Measure (FIM) is the most widely accepted functional assessment measure in use in the rehabilitation community. The FIM<sup>TM</sup> is an 18-item ordinal scale, used with all diagnoses within a rehabilitation population. It is viewed as most practical for assessment of progress during inpatient rehabilitation (State University of New York at Buffalo, 1997) and is assessed as part of normal rehabilitation care at admission and discharge from the rehabilitation unit. FIM<sup>TM</sup> efficiency is simply the change in FIM<sup>TM</sup> score divided by the length of rehabilitation stay and is used as marker of relative speed of functional change. We will evaluate for effects on both FIM<sup>TM</sup> motor and FIM<sup>TM</sup> cognitive scores.
- Symbol Digit Modalities Test[43]: The SDMT is a pencil and paper test for attention that takes approximately five minutes to administer and is frequently used in evaluations after TBI (DeMonte,

- 2009)) (Kalmar K, 2008) (Hanks R, 2008). The SDMT will be administered at enrollment and after intervention. The Interagency Workgroup on TBI Outcomes selected the Symbol Digit Modalities Test as CORE common data elements in TBI outcomes research.
- Positive and Negative Affect Schedule: The 20-item Positive and Negative Affect Schedule (PANAS), developed with a sample of undergraduate students and validated with adult populations, comprises two mood scales, one measuring positive affect and the other measuring negative affect. Each item is rated on a 5-point scale ranging from 1 = very slightly or not at all to 5 = extremely to indicate the extent to which the respondent has felt this way in the indicated time frame. This scale is used to measure affect over a range of times including: at this moment, today, the past few days, the past week, the past few weeks, the past year, and generally (on average). Watson et al. (Watson, 1988) reported Cronbach's alpha coefficients for the various time reference periods ranging from .86 to .90 for the Positive Affect scale and .84 to .87 for the Negative Affect scale. For the general period, alpha was.88 for Positive Affect and .87 for Negative Affect. Test-retest correlations for an 8-week period ranged from .47 to .68 for Positive Affect, .39 to .71 for Negative Affect (for the general time period, Positive Affect stability = .68, Negative Affect Stability = .71[44]).
- Therapy Participation: Participation in rehabilitation therapies will be evaluated at enrollment and again after light therapy (day 13) by the subject's therapist using a 0-100 scale of cooperation with therapy that has been previously utilized in this population.[45]
- Karolinska Sleepiness Scale (KSS): The KSS is a well-validated, widely used single question survey that examines current sleepiness.
- Barrow Neurological Institute Fatigue Scale (BNI-FS): The BNI-FS is a scale that was designed to examine fatigue during acute recovery from TBI. It has good internal consistency and appears to specifically examine a single psychometric construct of fatigue in patients with TBI (Wäljas M, 2012).
- Clinician Feasibility Survey: This is a likert scale survey to assess phototherapy intervention for ease of use, perceived relevance to rehabilitation care, and impression of effectiveness. This survey will be available in paper and electronic versions.

#### **XI.** Study Procedures:

#### **Screening and Enrollment:**

Patients' medical records will be screened for inclusion/exclusion criteria. Informed consent will be obtained from the subjects after they have been determined to be cognitively capable to consent for the study. A subject will be considered unable to give independent consent if they are still in PTA (as measured by the Galveston Orientation & Amnesia Test (GOAT), with a score <76) or their medical record at the time of enrollment specifies that they are unable for other reasons to independently consent. If a subject is unable to consider consent independently, proxy consent will be obtained from the legally authorized representative (LAR). This process is part of obtaining informed consent for the TBI Model System study. In addition, clinical staff and research staff have established communication lines to approach patients at appropriate times that do not interfere with patient clinical care.

#### **Baseline and Randomization:**

**Day 0-1** (2 days): After determining eligibility, the participant will be fitted with an Actiwatch (actigraphy) for continuous monitoring of activity levels both during the day and night (American Sleep Disorders Associatio, 1995). The Actiwatch will be worn continuously (with removal as needed for hygiene, shower or other clinical care) from enrollment to outcome measurement. Actiwatches will be fully charged and cleared of all previous data before being provided to a subject. Units will be set to record activity data in 60-second epochs. Actiwatches have sufficient built-in memory capacity and battery life to be used for approximately 30 days without recharging. Additionally, sleep logs that rate patient sleep are filled out every hour, between the hours of 2200-0600, this information is then obtained

as completion of the Makley scale. A complete review of symptoms and medical history will be obtained from the subject, LAR, and medical records.

**Day 2**: Baseline data collection is obtained (See Appendix for Baseline Data Collection Forms). Measures collected include: Symbol Digit Modalities Test, Positive and Negative Affect Schedule (PANAS), Barrow Neurological Fatigue Scale. Clinical Staff, will be asked if there was sleep difficulties and therapist will be asked to rate therapy participation for that day.

**Day 2:** Randomization. After baseline testing is completed, subjects will be randomized (50:50) using a 2-level stratification design based on two pieces of information:

- 1) Center (U. Washington-Seattle, Baylor-Dallas, Mount Sinai-New York) and
- 2) Severity of Sleep Disturbance using Delirium Rating Scale-Revised 98 Item 1

The rating for the Delirium Rating Scale Item 1 are: 1=Mild, 2=Moderate, 3=Severe (Nakase-Richardson R S. M., Prospective evaluation of the nature, course, and impact of acute sleep abnormality following TBI, 2013) Using an Access Database, developed by Jason Barber at the University of Washington, centers will randomize the participant into either the Bright White Light Group or the Dim Red Light Group. [46]

#### **Light Therapy:**

Days 3-13: Each morning for 10 days, the research and/or nursing staff will set up the Litebook® device in the marked out area of the bedside table. The light will be between 12 and 24 inches from the subject, allowing light to reach the subject's eyes. The subject will be in front of the device for 30 minutes, eating or otherwise doing relaxing activities and will have the eyes open. Both BWL and RL will be delivered using a Litebook® (The Litebook Company Ltd; Medicine Hat, Alberta, Canada). The Litebook® is a small (6 inch x 5 inch x 1 inch) unit with an attached stand that is placed 12-24 inches from the user's face and within 45 degrees of the visual field per manufacture guidance. Both the BWL and RL devices contain a data log to track the times at which the light box is turned off and on allowing the total time of exposure to be calculated. The cases for the BWL and RL units are visually identical. Research Staff will setup the Litebook ® on the bedside/over bed table as part of the subjects' morning/breakfast daily routine. The research staff will check in with nursing staff and the patient/LAR regarding adverse effects each day. Study medical staff will also be available for study questions or problems at other times and the patient's primary medical service will also be following for their overall medical care per routine. Nursing staff will be trained regarding the light exposure protocol as part of preparation for the study and the individualized setup for each subject will be reviewed and diagrammed in their room on enrollment. Subjects will receive 10 morning sessions of their assigned light therapy (BWL vs. RL).

#### **Additional Data Collected**

- 1) Sleep Logs: Sleep logs will be integrated with overnight nursing rounds. Trained nursing staff will perform regular ratings every hour of sleep/wakefulness between 2200-0600 using the Makley Scale, a 4-point ordinal scale ranging from 0 (asleep) to 3 (awake). This paper sleep log will be collected daily by the research study staff. This is part of routine rehabilitation care and will not add any sleep disruption for study participants. Sleep logs will be used as one tool to help interpret overall actigraphy data patterns during analysis.
- 2) Therapy Participation: The physical therapist will be asked by the research staff to rate at both baseline days and on the final two days outcome assessment time points.
- 3) Clinical Staff feedback: phototherapy intervention will rated using a likert scale on the following categories:

- a. Ease of use
- b. Perceived relevance to rehabilitation care
- c. Impression of effectiveness.

## **Post Light Therapy Outcome Assessment**

**Day 13**: At the conclusion of the light therapy sessions (and prior to discharge from rehabilitation), a blinded Outcomes Examiner will complete the post therapy outcome assessment. This assessment will include the following:

- Symbol Digit Modalities Test
- o Positive and Negative Affect Schedule (PANAS)
- o Barrow Neurological Fatigue Scale

#### XII. Data Analysis

The primary outcome is the between-group difference (BWL vs. RL exposure) in average sleep efficiency at baseline compared to after 10 days of light treatment. ANOVA will be used to compare groups controlling for demographics, injury severity, and use of medications.

Secondary outcomes (mood, therapy participation, attention, daytime sleepiness/fatigue) between groups assessed at baseline and after 10 days of light therapy will be compared using repeated measures ANOVA. FIM<sup>TM</sup> efficiency and inpatient rehabilitation length of stay will also be compared between groups using ANOVA controlling for the same variables as the primary outcome. Descriptive analysis will summarize responses to the nursing burden questions including estimated staff time for the intervention.

Initial scoring of the data will be done by each participating site with Actiware 5, a computer program which uses validated algorithms to determine whether an epoch of activity is "sleep" or "wake". The Actiware 5 software calculates sleep/wake statistics based on night intervals and provides these statistics for each interval (night), as well as a mean of all intervals (nights). Using a set interval of sleep, the software scores each epoch (minute) as sleep or wake, based on a specific internal algorithm and provides analysis of data, including sleep onset latency, sleep efficiency, sleep time, wake time, % sleep, % wake, naps, resting and normal night time sleep. The Actigraphy software does not provide circadian activity rhythms analysis. The raw, de-identified actigraphy data will be transmitted in an encrypted zip file via email to the NDSC and stored on a secure server for further analyses. Dr. Fogelberg will export edited epoch-by-epoch activity data to SAS programs to perform standard circadian activity analysis including calculation of Amplitude, Acrophase, Mesor, and the F-statistic. The activity level per epoch (minute) is used to estimate circadian activity rhythms. Circadian activity rhythms are analyzed by fitting each subject's activity data to a 5-parameter extended cosine model.

## XIII. Data Management

Table 2. Performance measures.

| Performance Area | Goal | Review<br>Schedule | <b>Evaluation Method</b> | Accountability* |
|---|---|---|---|---|
| <b>Pre Enrollment Activitie</b> | S | | | |
| Manual of Procedures | | | Ready for IRB | Glorieux, Bell,<br>Hoffman |
| IRB Submission | | | IRB approval | Glorieux,<br>Hoffman, Dubiel |
| Database complete | | | Trial data entry | Glorieux, Barber,<br>NDSC |
| Actigraphic data handling plan complete | | | Protocol | Fogelberg |
| Research Assistant trained | | | Observation of test administration and scoring, physical set-up | Glorieux,<br>Zumsteg, Dubiel |
| <b>Study Binders</b> | | | | Wasmund |
| Investigator | | | | Wasmund, |
| Communication | | | | Glorieux,<br>Zumsteg, Hoffman |
| Post-Enrollment Activiti | es | | | ζ, |
| <b>Enrollment per month</b> | | | Enrollment report | Glorieux |
| <b>Completion of</b> | | Monthly | Review by PI, | Wasmund, Site |
| baseline assessments | | | Data Report | Coordinators |
| <b>Completion of</b> | | Monthly | Review by PI, | Wasmund, Site |
| intervention | | | Data Report | Coordinators |
| <b>Completion of outcome</b> | | Quarterly | Review by PI, | Glorieux, Site |
| assessments | | _ | Data Report | Coordinators |
| Data Safety<br>Monitoring | 100% | Quarterly<br>and as<br>needed | Review by PI, Quarterly report to Medical Monitor | Olson, Hoffman,<br>Zumsteg |
| Data audit | 95% agreement | Quarterly | Rescoring and coding of 5% of assessments | Glorieux |
| Data Analysis/Dissemina | tion | | | |
| Complete Data<br>Analysis | | | | Hoffman, Dubiel,<br>Zumsteg,<br>Fogelberg |
| Complete primary report of study | | | Submission of manuscript for review | Hoffman et al |
| Design next study | | | Submission of | Investigators |

| grant proposal | 1 |
|----------------|---|
| grani proposai | i |
| 0 pp | |

#### **Identifiers**

Each study site will have specific site ID numbers; subjects will be assigned a unique number in consecutive order with site identification. These numbers will be assigned locally using the TWILIGHT Study Access Database. Study number, rather than name or medical record, will be on data collection forms. Consent forms with identifying information and contact forms will be filed separately from other study material and will be kept in a secure location (locked file or secure, password protected file on secure server, also with password protection). The link between study and identifying data will be destroyed as specified in the site's IRB documents.

## **Confidentiality**

Hard copies of study files will be kept in a locked cabinet or a secure location accessible only to individuals who have signed institutional confidentiality agreements. Study number will be on data collection forms (other than the locator form with contact information). Data in electronic form will be encrypted and stored on a University of Washington or NIDRR server only accessible by authorized personnel. Identified information such as name, address, medical record number or phone numbers needed to initially identify participants or their LAR will be kept in separate files from the study data.

Only study personnel as well as representatives of the human protection offices, and representatives of the funding agency will have access to study records. The study will not intentionally collect any data that would need to be shared with state or local authorities. If the participant responds to assessment items or volunteers information about an intent to harm themselves or others (such as in review of systems questions), a standard IRB approved protocol (identical to the TBI Model System protocol) will be executed to manage such disclosures to ensure participant or others' safety and the subject's inpatient rehabilitation resident or attending physician will be informed verbally immediately.

## Disposition of data

At each study site hard copy data will be stored in locked file cabinets or a secure location while the study is ongoing. When the study is complete, the data will be sent to a secure institutional records management location at each site similar to those used to store archived medical records as required by local and other regulations as applicable to each site. Washington State law requires clinical trial data be retained for 25 years. Electronic data will be entered into a database developed by the National Data and Statistical Center using an ACCESS database that will be kept behind secure firewall on servers accessible to site data managers with password-protected access. At the end of the study, each investigator will get a copy of the de-identified data. At the end of the study, all local copies of the contact information files will be destroyed.

**ACG data:** De-identified actigraphic data will be transmitted in an encrypted ZIP file via UW secure and government email to the NDSC and stored on a secure, password-protected server accessible only to site data managers and PIs.

Demographic, Injury Characterization, Traumatic Brain Injury Model System (TBIMS)

**Outcomes:** Data will be recorded on paper or directly into database developed by the National Data and Statistical Center at Craig Hospital using an ACCESS database that will be kept behind secure firewall on servers accessible to site data managers with password-protected access. Hard copies of the data will be stored in locked file cabinets or a secure location while the study is ongoing. Only de-identified data is released from the NDSC.

**Paper and Pencil Tests, Cognitive Tests, Interviews:** Data will be recorded on paper. All subjective questionnaires and cognitive testing scores will be entered into the secure database developed by the TBIMS NDSC at Craig Hospital using an ACCESS database that will be kept behind secure firewall on servers accessible to site data managers with password-protected access. Hard copies of the data will be stored in locked file cabinets or a secure location while the study is ongoing.

## **Sharing study results**

Treatment conducted as part of this study may be of benefit to an individual participant (e.g. progress on cognitive testing over time). The main sharing of study results, however, will be with the general public and medical community which may benefit from our study outcome. We plan to report our findings in published material and at medical conferences. Data sharing will follow the TBIMS protocol.

### XIV. Safety and Adverse Events

Each subject will be followed medically daily by their rehabilitation resident and attending physicians and have 24 hour monitoring by rehabilitation nursing. The research assistant at each site will check in with the patient/LAR and nursing staff daily Monday through Friday to elicit any concerns. Jared Olson, M.D. a physiatrist in the University of Washington's Department of Rehabilitation Medicine has expertise in TBI treatment and research procedures and has agreed to be the Data Safety Monitor (DSM). He will receive a quarterly summary of all Adverse Events for review and will be contacted by the study team within 24 hours of any Serious Adverse Event to review with the study physician. Any serious adverse event will be reported to the Human Subjects Division as well immediately. At quarterly intervals after subject enrollment begins, the DSM will review and evaluate the studies' clinical efficacy and safety data. The DSM will monitor study progress, examine adverse events (AEs) and serious adverse events (SAEs), and recommend the continuation without change, suspension, or termination of a study.

#### XV. Definitions

#### **Unanticipated Problems Involving Risk to Subjects or Others**

Any incident, experience, or outcome that meets all of the following criteria:

- <u>Unexpected in nature, severity, or frequency</u> (i.e. not described in study-related documents such as the IRB-approved protocol or consent form, the investigators brochure, etc)
- Related or possibly related to participation in the research (i.e. possibly related means there is a reasonable possibility that the incident experience, or outcome may have been caused by the procedures involved in the research)
- <u>Suggests that the research places subjects or others at greater risk of harm</u> (including physical, psychological, economic, or social harm).

Rev: 9/2/2014

#### **Adverse Event**

An *adverse event* (AE) is any symptom, sign, illness or experience that develops or worsens in severity during the course of the study. Intercurrent illnesses or injuries should be regarded as adverse events. Abnormal results of diagnostic procedures are considered to be adverse events if the abnormality results in study withdrawal, is associated with a serious adverse event, is associated with clinical signs or symptoms, or is considered by the investigator to be of clinical significance.

#### **Serious Adverse Event**

Adverse events are classified as serious or non-serious. A *serious adverse event* is any AE that is: fatal, life-threatening, prolongs hospital stay, results in persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event.

All adverse events that do not meet any of the criteria for serious should be regarded as **non-serious adverse event.** 

**Important medical events** are those that may not be immediately life threatening, but are clearly of major clinical significance. They may jeopardize the subject, and may require intervention to prevent one of the other serious outcomes noted above.

## **Adverse Event Reporting Period**

The study period during which adverse events must be reported is normally defined as the period from the initiation of any study procedures to the end of the study treatment follow-up. For this study, the study treatment follow-up is defined as 2 days following the last study treatment (Day 15).

### Hospitalization

Subjects will be hospitalized patients receiving care for their recent traumatic brain injury. Therefore, hospitalization is a requirement to be a part of this study, and will not be included as an adverse event for this study.

## XVI. Recording of Adverse Events

At each contact with the subject, the study staff must seek information on adverse events by specific questioning. Information on all adverse events should be recorded immediately in the source document, and also in the appropriate adverse event module of the case report form (CRF). All clearly related signs, symptoms, and abnormal diagnostic procedures results should recorded in the source document, though should be grouped under one diagnosis.

All adverse events occurring during the study period must be recorded. The clinical course of each event should be followed until resolution, stabilization, or until it has been determined that the study treatment or participation is not the cause. Serious adverse events that are still ongoing at the end of the study period must be followed up to determine the final outcome. Any serious adverse event that occurs after the study period and is considered to be possibly related to the study treatment or study participation should be recorded and reported immediately.

Minimum information required for each AE includes type of event, duration (start and end dates), severity, seriousness, causality to study, action taken, and outcome.

## **Evaluating Adverse Events**

Assessment should include the intensity (severity) of the event and the relationship to Study Intervention(s).

Severity of AEs will be graded by the Investigator using the following criteria as guidelines:

- 1) *Mild*: Nuisance, barely noticeable.
- 2) *Moderate:* Uncomfortable, troublesome symptoms not significantly interfering with daily activities or sleep.
- 3) **Severe:** Symptoms significantly interfere with daily activities or sleep.

The <u>relationship of the AE to the study treatment</u> should be specified by the Investigator, using the following definitions:

1) Not Related: Concomitant illness, accident or event with no reasonable association with treatment.

- 2) *Unlikely*: The reaction has little or no temporal sequence from administration of the study treatment, and/or a more likely alternative etiology exists.
- 3) *Possibly Related*: The reaction follows a reasonably temporal sequence from administration of the treatment and follows a known response pattern to the suspected treatment; the reaction could have been produced by the study treatment or could have been produced by the subject's clinical state or by other modes of therapy administered to the subject.
- 4) *Probably Related*: The reaction follows a reasonable temporal sequence from administration of study treatment; is confirmed by discontinuation of the study treatment or by rechallenge; and cannot be reasonably explained by the known characteristics of the subject's clinical state.
- 5) **Definitely Related**: The reaction follows a reasonable temporal sequence from administration of study treatment; that follows a known or expected response pattern to the study treatment; and that is confirmed by improvement on stopping or reducing the dosage of the study treatment, and reappearance of the reaction on repeated exposure.

## **Notifying the Principal Investigator**

Any study-related unanticipated problem posing risk of harm to subjects or others that are not Adverse Events should be reported on the "*Unanticipated Problems Form*". Any type of serious adverse event, must be reported to the site Principal Investigator or designee within 1 business day of the event. Within the following 48 hours, the investigators must provide further information on the serious adverse event or the unanticipated problem in the form of a written narrative. This should include a copy of the completed Serious Adverse Event form, and any other diagnostic information that will assist the understanding of the event.

#### **Notifying the Local IRB**

At the University of Washington, Dr. Jeanne Hoffman or Dr. Jennifer Zumsteg will be responsible for safety reporting to the IRB and complying with their reporting requirements. The other sites for this project will have an investigator who is responsible for safety reporting to their local IRBs. Copies of each report and documentation of IRB notification and receipt will be kept in the locked secured study file.

## **Notifying the Data Safety Monitor**

Unanticipated problems posing risks to subjects or others and serious adverse events associated with the research will be forwarded to the Data Safety Monitor of the study at the University of Washington, within 24 hours.

## Stopping Rules

There are no planned interim or futility analyses. The Data Safety Monitor may recommend stopping for safety based on overall study review.

## **Independent Data Safety Monitor**

The Data Safety Monitor is required to review all unanticipated problems involving risk to volunteers or others, serious adverse events and all volunteer deaths associated with the protocol and provide an unbiased written report. At a minimum the Data Safety Monitor should comment on the outcomes of the event or problem and in the case of a serious adverse event or death comment on the relationship to participation in the study. The Data Safety Monitor should also indicate whether he concurs with the details of the report provided by the study investigator.

#### XVII. Ethical Considerations/Protection of Human Subjects

Ethical Conduct of the Study

This study is to be conducted according to US and international standards of Good Clinical Practice (FDA Title 21 part 312 and International Conference on Harmonization guidelines), applicable government regulations and Institutional research policies and procedures.

#### Institutional Review Board (IRB)

This protocol and any amendments will be submitted to a properly constituted Institutional Review Board (IRB), in agreement with local legal prescriptions, for formal approval of the study conduct. The decision of the IRB concerning the conduct of the study will be made in writing to the investigator.

#### Subject Information and Informed Consent

This study will be conducted in compliance with Title 45 Part 46 of the CFR pertaining to informed consent. At the first visit, subjects will give their written consent to participate in the study after having been informed about the nature and purpose of the study, participation/termination conditions, risks, and potential benefits. Informed consent is a process that is initiated prior to the individual's or proxy's agreeing to participate in the study and continuing throughout the individual's study participation. Extensive discussion of risks and possible benefits of this therapy will be provided to the participants and their families. Consent forms describing in detail the Study Agent(s)/Intervention(s) study procedures and risks are given to the participant/proxy and written documentation of informed consent is required prior to starting study agent/intervention. Consent forms will be IRB approved and the participant/proxy will be asked to read and review the document. Upon reviewing the document, the investigator will explain the research study to the participant/proxy and answer any questions that may arise. The participants/proxies should have sufficient opportunity to discuss the study and process the information in the consent process prior to agreeing to participate. The participants/proxies may withdraw consent at any time throughout the course of the study. A copy of the informed consent document will be given to the participants/proxies for their records. The rights and welfare of the participants will be protected by emphasizing to them that the quality of their medical care will not be adversely affected if they decline to participate in this study.

## Sample Characteristics that Raise Special Concerns

Participants may not be sufficiently able to independently provide informed consent. We will have proxy consent forms for the subject and the Legally Authorized Representative (LAR) in this case. Decision making capacity assessment is described in the above study procedure narrative. We do not anticipate re-consenting subjects as the study duration is only 10 days of intervention.

# XVIII. Potential Risks, Potential Benefits, Intent to Benefit, and Risk/Benefit Ratio Potential risks

Subjects may experience an adverse reaction to the active or comparison treatment; significant adverse reactions are unlikely given literature on these light therapy interventions in a variety of populations. The intervention involves exposure to light, which can be bright and which some participants may find bothersome. Side effects of the bright white light are generally mild and subside but can include hypomania, irritability, headache, nausea, eye strain or vision changes and sleep changes (Chang AM, 2012). Other side effects are not anticipated given the study target population and the study team's experience with sleep changes after TBI and light therapy. Other study procedures including the questions about cognition such as memory may be uncomfortable either physically or emotionally and will be approached respectfully and confidentially. The placement of the Actiwatch on the wrist will result in contact with the skin, and like any watch, could result in contact dermatitis. Contact Dermatitis is readily treated with skin lotion and may involve repositioning the device. Prior studies have not reported this as a problem.

As with any study, there is also a remote chance that an outside party may discover a participant's identity and participation in the study. Risk of physical harm or injury is unlikely given the mild nature of reported side effects in the literature regarding light exposure and the non-invasive nature of actigraphy. No risk to study personnel is anticipated.

Alternative common treatments for insomnia include sedative drugs / sleep medications, behavioral interventions and environmental modifications. These other interventions will be recorded and will not be blocked during this study.

## **Protection Against Risk**

- 1. We will have a Data Safety Monitor who is independent of the study to review regular reports of any reported related or unrelated adverse events as noted above. All serious adverse events will be reported within 24 hours to him as well as to the IRB, Dr. Hoffman and site PIs. Our DSM will be able to halt recruitment until any adverse events are thoroughly explored. A summary of all adverse events will be generated quarterly.
- 2. Subjects will be interviewed in private settings, will be counseled that they may refuse to answer any question, and will be reassured that the information they provide is confidential.
- 3. We will take all the usual steps to protect the confidentiality of personal information, including but not limited to dissociating identifying information from research data; using unique alpha-number coding systems that permit linkages to identifying data only via files that are stored separately; storage of data on password protected servers or computers; storage of paper data forms in locked files within locked rooms with access limited to approved research staff. All investigators and research staff are required to undergo HIPAA training and to sign a confidentiality agreement under the authority of the Human Subjects Division of the University of Washington and participating sites.

## Risk Management

Loss of Confidentiality: All of the paper-based assessments will be kept in locked file cabinets at the study site. All data will be identified by a subject number. The link between participant identities and subject number will be kept separately from the study data. All personnel will receive HIPAA training as required by the University of Washington's Human Subjects Division.

#### XIX. Importance of Knowledge to be Gained

At the completion of this study, we will have evidence on whether Bright White Light Therapy improves sleep after TBI. If this study is successful, we will have an **immediately available**, **effective**, **non-invasive** way of improving sleep for patients who have experienced a TBI that will enhance not only sleep timing but also thinking abilities and possibly long-term recovery after TBI.

#### **XX.** Study Finances

#### **Funding Source**

This study is financed through TBI Model System Grant for the 2012-2017 Grant Cycle. This a module multi-site project that will be conducted at three locations. All participating sites have received funding from the National Institute on Disability and Rehabilitation Research.

## Subject Stipends or Payments

There is no compensation planned for subjects who choose to participate in this study.

#### **XXI.** Overall Project Evaluation

Overall study data completeness, timeliness, and quality will be monitored by the study investigators. Automated data reports will be generated monthly, displaying information relevant to the milestones described in the previous section. For example, cumulative subject accrual rates, subject retention rates, inter-rater reliability, and data accuracy reports will be generated routinely to monitor progress toward goals. Progress toward study milestone will be discussed at the project meetings. Quarterly reports will be filed with the NIDRR project officer. Quarterly safety reports will be submitted to Dr. Olson. Annual reports will be filed with the TBIMS Annual Reports.

Investigators and key study personnel will meet by telephone bi-weekly prior to the initiation of the intervention to discuss progress. Investigators will meet twice yearly at the TBIMS Project Directors meeting. Site teams will meet weekly during the intervention period to discuss progress and barriers. If problems arise or tasks are not progressing as planned, Dr. Hoffman will work with the research team to devise an action plan. Plans will be put in writing with a timeline to correct the problem. Ms. Glorieux will track and follow-up on these plans. Any significant problems that would affect overall project outcomes will be reviewed with the NIDRR project officer to obtain additional assistance in developing an action plan.

**Table 3: Timeline of Research Activities** 

| | 2013 | 3 | 201 | 4 | 201 | 5 | 201 | 6 | 201 | 7 |
|---|---|---|---|---|---|---|---|---|---|---|
| Pre-Enrollment Activities | | | | | | | | | | |
| Complete feasibility study | X | | | | | | | | | |
| Manual of Procedures | X | | | | | | | | | |
| Primary site IRB | X | | | | | | | | | |
| Collaborator sites IRB | | X | | | | | | | | |
| Research Assistant Training | | X | | | | | | | | |
| Rehab Staff Training | | X | | | | | | | | |
| Post-Enrollment Activities | | | | | | | | | | |
| Cumulative Enrollment Target | | | | 43 | | 86 | | 128 | | |
| Data collection | | | X | X | X | X | X | X | | |
| Actigraphy interpretation | | | X | X | X | X | X | X | | |
| Data Analysis/Dissemination | | | | | | | | | | |
| Primary study report | | | | | | | | | X | |
| Manuscript preparation | | | | | | | | | X | X |

Figure 2. Project Staff Flow Chart

## List of Acronyms and Abbreviations

- **ACG** = Actigraphy
- **AE**= adverse event
- **BMI** = body mass index
- **BNI-FS** = Barrow Neurological Institute Fatigue Scale
- **BWL** = Bright white light (experimental treatment condition in this study)
- **DSM** = Data safety monitor
- GCS = Glasgow Coma Scale
- **GOAT** = Galveston Orientation and Amnesia Test
- **KSS** = Karolinska Sleepiness Scale
- LAR = Legally authorized representative
- NDSC = National Data and Statistical Center for the Traumatic Brain Injury Model S
- **NIDRR** = National Institute on Disability and Rehabilitation Research
- **PANAS** = Positive and Negative Affective Schedule
- **PTA** = Post-traumatic amnesia
- **RL** = Dim red light (comparison treatment condition in this study)
- SAE = Serious adverse event
- **SDMT** = Symbol Digit Modalities Test
- **TBI** = Traumatic brain injury
- **TBIMS** = Traumatic brain injury Model System

#### Works Cited

- 1. Orff, H.J., L. Ayalon, and S.P. Drummond, *Traumatic brain injury and sleep disturbance: a review of current research*, in *J Head Trauma Rehabil*. 2009: United States. p. 155-65.
- 2. Mathias JL, A.P., *Prevalence of sleep disturbances, disorders, and problems following traumatic brain injury: A meta analysis.* . Sleep Med, 2012;13: p. 898-905.
- 3. Ouellet, M.C., J. Savard, and C.M. Morin, *Insomnia following traumatic brain injury: a review*. Neurorehabil Neural Repair, 2004. **18**(4): p. 187-98.
- 4. Ouellet, M.C., S. Beaulieu-Bonneau, and C.M. Morin, *Insomnia in patients with traumatic brain injury: frequency, characteristics, and risk factors.* J Head Trauma Rehabil, 2006. **21**(3): p. 199-212.
- 5. Verma, A., V. Anand, and N.P. Verma, *Sleep disorders in chronic traumatic brain injury*. J Clin Sleep Med, 2007. **3**(4): p. 357-62.
- 6. Ayalon, L., et al., *Circadian rhythm sleep disorders following mild traumatic brain injury*. Neurology, 2007. **68**(14): p. 1136-40.
- 7. Makley, M.J., et al., *Prevalence of sleep disturbance in closed head injury patients in a rehabilitation unit*, in *Neurorehabil Neural Repair*. 2008: United States. p. 341-7.
- 8. Ohayon, M.M. and C.F. Reynolds, 3rd, *Epidemiological and clinical relevance of insomnia diagnosis algorithms according to the DSM-IV and the International Classification of Sleep Disorders (ICSD)*, in *Sleep Med.* 2009: Netherlands. p. 952-60.
- 9. Larson, E.B. and F.S. Zollman, *The effect of sleep medications on cognitive recovery from traumatic brain injury.* J Head Trauma Rehabil, 2010. **25**(1): p. 61-7.
- 10. Flanagan, S.R., B. Greenwald, and S. Wieber, *Pharmacological treatment of insomnia for individuals with brain injury*, in *J Head Trauma Rehabil*. 2007: United States. p. 67-70.
- 11. Carter, K.A., C.J. Lettieri, and J.M. Pena, *An unusual cause of insomnia following IED-induced traumatic brain injury*. J Clin Sleep Med, 2010. **6**(2): p. 205-6.
- 12. Chesson, A.L., Jr., et al., *Practice parameters for the use of light therapy in the treatment of sleep disorders. Standards of Practice Committee, American Academy of Sleep Medicine.* Sleep, 1999. **22**(5): p. 641-60.
- 13. Englander, J., et al., *Fatigue after traumatic brain injury: Association with neuroendocrine, sleep, depression and other factors.* Brain Inj, 2010. **24**(12): p. 1379-88.
- 14. Banks, S. and D.F. Dinges, *Behavioral and physiological consequences of sleep restriction*. J Clin Sleep Med, 2007. **3**(5): p. 519-28.
- 15. Mishima, K., et al., Morning bright light therapy for sleep and behavior disorders in elderly patients with dementia. Acta Psychiatr Scand, 1994. **89**(1): p. 1-7.
- 16. Riemersma-van der Lek, R.F., et al., *Effect of bright light and melatonin on cognitive and noncognitive function in elderly residents of group care facilities: a randomized controlled trial.* JAMA, 2008. **299**(22): p. 2642-55.
- 17. Fogelberg, D.J., et al., Association of sleep and co-occurring psychological conditions at 1 year after traumatic brain injury. Arch Phys Med Rehabil, 2012. **93**(8): p. 1313-8.
- 18. Reeves, G.M., et al., *Improvement in depression scores after 1 hour of light therapy treatment in patients with seasonal affective disorder*, in *J Nerv Ment Dis.* 2012: United States. p. 51-5.
- 19. Chang, A.M., et al., *Human responses to bright light of different durations*, in *J Physiol*. 2012: England. p. 3103-12.
- 20. Riemersma-van der Lek, R.F., et al., *Effect of bright light and melatonin on cognitive and noncognitive function in elderly residents of group care facilities: a randomized controlled trial*, in *JAMA*. 2008: United States. p. 2642-55.
- 21. Terman, M. and J.S. Terman, *Light therapy for seasonal and nonseasonal depression: efficacy, protocol, safety, and side effects.* CNS Spectr, 2005. **10**(8): p. 647-63; quiz 672.

- 22. Wirz-Justice, A. and M. Terman, *Chronotherapeutics (light and wake therapy) as a class of interventions for affective disorders*, in *Handb Clin Neurol*. 2012: Netherlands. p. 697-713.
- 23. Morgenthaler, T.I., et al., *Practice parameters for the clinical evaluation and treatment of circadian rhythm sleep disorders. An American Academy of Sleep Medicine report.* Sleep, 2007. **30**(11): p. 1445-59.
- 24. Zollman, F.S., C. Cyborski, and S.A. Duraski, *Actigraphy for assessment of sleep in traumatic brain injury: case series, review of the literature and proposed criteria for use.* Brain Inj, 2010. **24**(5): p. 748-54.
- 25. Ayalon, L., et al., *Circadian rhythm sleep disorders following mild traumatic brain injury*, in *Neurology*. 2007: United States. p. 1136-40.
- 26. Fogelberg, D.J., et al., Association of sleep and co-occurring psychological conditions at 1 year after traumatic brain injury, in Arch Phys Med Rehabil. 2012, 2012 American Congress of Rehabilitation Medicine. Published by Elsevier Inc: United States. p. 1313-8.
- 27. Watson, N.F., et al., *Hypersomnia following traumatic brain injury*. J Clin Sleep Med, 2007. **3**(4): p. 363-8.
- 28. Gumber, S., et al., *Treatment of post TBI fatigue with light exposure*, in *American Psychological Association*, *Division of Rehabilitation Psychology 15th Annual Congress*. 2013: Jacksonville, FL.
- 29. Wood, R.L., et al., *Clinical and cost effectiveness of post-acute neurobehavioural rehabilitation*. Brain Inj, 1999. **13**(2): p. 69-88.
- Whitmore, R.G., et al., *Is aggressive treatment of traumatic brain injury cost-effective?* J Neurosurg, 2012. **116**(5): p. 1106-13.
- 31. Jason M. Sutherland, P.D., Elliott S. Fisher, M.D., M.P.H., and Jonathan S. Skinner, Ph.D., *Getting Past Denial The High Cost of Health Care in the United States*. NEJM, 2009. **361**(13): p. 1227-1230.
- 32. Cuthbert JP, C.J., Whiteneck GG, Harrison-Felix C, Graham JE, Bell JM et al., *Extension of the representativeness of the Traumatic Brain Injury Model Systems National Database: 2001 to 2010.* J Head Trauma Rehabil. United States, 2012: p. E15-27.
- 33. Lakshmanan, R., Loo, J. A., Drake, T., Leblanc, J., et al., *Metabolic crisis after traumatic brain injury is associated with a novel microdialysis proteome*. Neurocrit Care 2010: p. 12, 324-336.
- 34. Zollman FS, L.E., Wasek-Throm LK, Cyborski CM, Bode RK., *Acupuncture for treatment of insomnia in patients with traumatic brain injury: a pilot intervention study.* J Head Trauma Rehabi, Mar-Apr 2012: p. 27(2):135-42.
- 35. Cuthbert, J.P., et al., *Extension of the representativeness of the Traumatic Brain Injury Model Systems National Database: 2001 to 2010*, in *J Head Trauma Rehabil.* 2012: United States. p. E15-27.
- 36. Netzer, N.C., et al., *Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome*, in *Ann Intern Med*. 1999: United States. p. 485-91.
- 37. Trzepacz PT, M.D., Torres R, Kanary K, Norton J, Jimerson N., *Validation of the Delirium Rating Scale Revised: Comparison with the Delirium Rating Scale and the Cognitive Test for Delirium.* J Neuropsychiatr Clin Neuroscience, 2001: p. 13:229-42.
- 38. Makley MJ, E.J., Drubach DA, Kreuz AJ, Celnik PA, Tarwater PM, *Prevalence of sleep disturbance in closed head injury patients in a rehabilitation uni*. Neurorehabil Neural Repair., 2008: p. 341-7.
- 39. *Guide for the Uniform Data Set for Medical Rehabilitation (including the FIM(TM) instrument.* 1997: Buffalo, NY 14214-3007, Buffalo, NY 14214-3007.
- 40. Shum D, M.K., Bain J., Construct validity of eight tests of attention: Comparison of normal and closed head injured samples. Clinical Neuropsychologist 1990: p. 4(2):151-62.
- 41. Watson, D., Clark, L. A., & Tellegen, A., *Development and validation of brief measures of positive and negative affect: The PANAS scales.* Journal of Personality and Social Psychology, 1988: p. 54 (6), 1063-1070.
- 42. Silva, M.A., et al., *Posttraumatic confusion predicts patient cooperation during traumatic brain injury rehabilitation.* Am J Phys Med Rehabil, 2012. **91**(10): p. 890-3.



#### I. References

- Genetic influences on outcome following traumatic brain injury. (2007). Neurochem Res, 32, 905-915.
- Abdullah, L. C. (2011). Proteomic CNS Profile of Delayed Cognitive Impairment in Mice Exposed to Gulf War Agents. *Neuromolecular Med*, 13, 275-288.
- Abdullah, L. E. (2012). Lipidomic Profiling of Phosphocholine Containing Brain Lipids in Mice with Sensorimotor Deficits and Anxiety-Like Features After Exposure to Gulf War Agents. *Neuromolecular Med*.
- Abdullah, L. L. (2009). Serum Abeta levels as predictors of conversion to mild cognitive impairment/Alzheimer disease in an ADAPT subcohort . *Mol Med* , 15, 432-437.
- Abdullah, L. L.-g. (2009). High serum Abeta and vascular risk factors in first-degree relatives of Alzheimer's disease patients. *Mol Med* , 15, 95-100.
- Abdullah, L. R. (2009). Proteomic Analysis of Human Neuronal Cells Treated with the Gulf War Agent Pyridostigmine Bromide. *J Proteomics Bioinform*, 2, 439-444.
- Ait-ghezala, G. A. (2008). Diagnostic utility of APOE, soluble CD40, CD40L, and Abeta1-40 levels in plasma in Alzheimer's disease. *Cytokine*, 44, 283-287.
- Ait-Ghezala, G. M. (2005). Genomic regulation after CD40 stimulation in microglia: relevance to Alzheimer's disease. *Brain Res Mol Brain Res*, 140, 73-85.
- Akerstedt T, G. M. (1990). Subjective and objective sleepiness in the active individual. *International Journal of Neuroscience*, 52: 29–37.
- Alger SE, L. H. (2012 Jun 23). Slow wave sleep during a daytime nap is necessary for protection from subsequent interference and long-term retention. . *Neurobiol Learn Mem*.
- American Sleep Disorders Associatio. (1995). Practice parameters for the use of actigraphy in the clinical assessment of sleep disorders. *Sleep*, 18:285-7.
- Ayalon L, B. K. (2007). Circadian rhythm sleep disorders following mild traumatic brain injury. *Neurology*, 1136-40.
- Banks S, D. D. (2007). Behavioral and physiological consequences of sleep restriction. *J Clin Sleep Med*, 3(5):519-28.
- Bennett, C. C. (1995). Evidence that the APOE locus influences rate of disease progression in late onset familial Alzheimer's Disease but is not causative. *Am J Med Genet*, 60, 1-6.
- Berson DM, D. F. (2002). Phototransduction by retinal ganglion cells that set the circadian clock. *Science*, 295(5557):1070-1073.
- Borgaro SR, G. S. (2004). Fatigue after brain injury: initial reliability study of the BNI Fatigue Scale. *Brain Inj*, 18:685-90.
- Cantor, J. B., Cicerone, K., Dijkers, M. P., Gordon, W., Hammond, F. M., Kolakowsky-Hayner, S. A., . . . Spielman, L. (2012). Insomnia, fatigue, and sleepiness in the first 2 years after traumatic brain injury: an NIDRR TBI model system module study. *The Journal of head trauma rehabilitation*, 27(6):E1-14.
- Carter KA, L. C. (2010). An unusual cause of insomnia following IED-induced traumatic brain injury. *J Clin Sleep Med*, 6(2):205-6.
- Castriotta RJ, A. S. (2009). Treatment of sleep disorders after traumatic brain injury. *J Clin Sleep Med*, 5:137-44
- Castriotta RJ, W. M. (June 15, 2007). Prevalence and consequences of sleep disorders in traumatic brain injury. *J CLin Sleep Med*, 349-56.
- Chang AM, S. N. (2012). Human responses to bright light of different durations. J Physiol, 590(Pt 13):3103-12.
- Chesson AL, J. L.-D. (1999). Practice parameters for the use of light therapy in the treatment of sleep disorders. Standards of Practice Committee, American Academy of Sleep Medicine. *Sleep*, 2.
- Chuang, P. C. (2010). Neuroglobin genetic polymorphisms and their relationship to functional outcomes after traumatic brain injury. *J Neurotrauma*, 27, 999-1006.
- Cole RJ, K. D. (1992). Automatic sleep/wake identification from wrist activity. Sleep, 15 (5):461–469.

- Crawford, F. A. (2000). Gender-specific association of the angiotensin converting enzyme gene with Alzheimer's diseas. *Neurosci Lett*, 280, 215-219.
- Crawford, F. C. (2000). A polymorphism in the cystatin C gene is a novel risk factor for late-onset Alzheimer's disease. *Neurology*, 55, 763-768.
- Crawford, F. C. (2000). The genetic association between Cathepsin D and Alzheimer's disease. *Neurosci Lett*, 289, 61-65.
- Crawford, F. C. (2006). Cocaine induced inflammatory response in human neuronal progenitor cells. *J Neurochem*, 97, 662-674.
- Crawford, F. C. (2012). Identification of plasma biomarkers of TBI outcome using proteomic approaches in an APOE mouse model. *J Neurotrauma*, 29, 246-260.
- Crawford, F. F. (1999). No genetic association between polymorphisms in the Tau gene and Alzheimer's disease in clinic or population based samples. *Neurosci Lett*, 266, 193-196.
- Crawford, F. T. (1999). The alpha-2 macroglobulin gene is not associated with Alzheimer's disease in a case-control sample. *Neurosci Lett*, 270, 133-136.
- Crawford, F. V. (2002). APOE genotypeinfluences acquisition and recall following traumatic brain injury. . *Neurology*, 58, 1115-1118.
- Crawford, F. W. (2009). Apolipoprotein E-genotype dependent hippocampal and cortical responses to traumatic brain injury. *Neuroscience*, 159, 1349-1362.
- Cuthbert JP, C. J.-F. (2012). Extension of the representativeness of the Traumatic Brain Injury Model Systems National Database: 2001 to 2010. . *J Head Trauma Rehabil. United States*, E15-27.
- Dardiotis, E. F. (2010). Genetic association studies in patients with traumatic brain injury. *Neurosurg Focus*, 28. Dash MB, C. C. (2009). Long-term homeostasis of extracellular glutamate in the rat cerebral cortex across sleep
- Dash MB, C. C. (2009). Long-term homeostasis of extracellular glutamate in the rat cerebral cortex across sleep and waking states. *J. Neuroscience*, 29:620-9.
- DeMonte, V. G. (2009)). Improved sensitivity of the rapid screen of mild traumatic brain injury. *J Clin Exp Neuropsychology*, 6, 1-11.
- Diaz-Arrastia, R. &. (2006). Genetic factors in outcome after traumatic brain injury: what the human genome project can teach us about brain trauma. *J Head Trauma Rehabil*, 361-374.
- Diekelmann S, W. I. (2009). The whats and whens of sleep-dependent memory consolidation. *Sleep Med Rev*, 13:309-21.
- DM, B. (2007). Phototransduction in ganglion-cell photoreceptors. *Pflugers Arch*, 454(5):849-855.
- Englander J, B. T. (2010). Fatigue after traumatic brain injury: Association with neuroendocrine, sleep, depression and other factors. *Brain Inj*, 24(12):1379-88.
- Ferguson, S. M. (2010). Apolipoprotein E genotype and oxidative stress response to traumatic brain injury. *Neuroscience*, 168, 811-819.
- Flanagan SR, G. B. (2007). Pharmacological treatment of insomnia for individuals with brain injury. *J Head Trauma Rehabil*, 67-70.
- Fogelberg DJ, H. J. (2012). Association of sleep and co-occurring psychological conditions at 1 year after traumatic brain injury. Fogelberg DJ, Hoffman JM, Dikmen S, Temkin NR, Bell KR. Association of sleep and co-occurring psychological conditions at 1 year after traumatic brain injury. Arch Phys Med Rehabil., 1313-8.
- Forbes D, C. I. (2011). Light therapy for managing cognitive, sleep, functional, behavioural, or psychiatric disturbances in dementia (Cochrane Database Syst Rev 2009). *Sleep*, 34:111-9.
- Freeman, T. R. (2005). Neuropsychiatric associations of apolipoprotein E alleles in subjects with combatrelated posttraumatic stress disorder. . J Neuropsychiatry Clin Neurosci, 17, 541-543.
- Friedman L, S. A.-I. (May 2012). Brief morning light treatment for sleep/wake disturbances in older memory-impaired individuals and their caregivers. *Sleep Med*, 13(5):546-9.
- Gao, W.-M. C. (2007). A gel-based proteomic comparison of human cerebrospinal fluid between inflicted and non-inflicted pediatric traumatic brain injury. *J Neurotrauma*, 24, 43-53.

- Genét, G. F. (2013). Trauma-induced coagulopathy: standard coagulation tests, biomarkers of coagulopathy, and endothelial damage in patients with traumatic brain injury. *J Neurotrauma*, 30, 301-306.
- Gong, D. H. (2012). Prognostic relevance of circulating endothelial progenitor cells for severe traumatic brain injury. *Brain Inj*, 26, 291-297.
- Gumber S, S. A. (2013). Treatment of post TBI fatigue with light exposure. Jacksonville, FL, United States: American Psychological Association, Division of Rehabilitation Psychology 15th Annual Congress.
- Hanks R, M. S.-R. (2008). The predictive validity of a brief neuropsychological battery for persons with traumatic brain injury. *Arch Phys Med Rehabil*, 89:950-7.
- Haqqani, A. H. (2007). Biomarkers and diagnosis; protein biomarkers in serum of pediatric patients with severe traumatic brain injury identified by ICAT-LC-MS/MS. *J Neurotrauma*, 24, 54-74.
- Hendoui, N. B. (2013). Reliability of calcium-binding protein S100B measurement toward optimization of hyperosmolal therapy in traumatic brain injury. *Eur Rev Med Pharmacol Sci*, 17, 477-485.
- Ho, L. Z.-O. (2012). Elevated plasma MCP-1 concentration following traumatic brain injury as a potential "predisposition" factor associated with an increased risk for subsequent development of Alzheimer's disease. *J Alzheimers Dis*, 31, 301-313.
- Irizarry, M. (2004). Biomarkers of Alzheimer disease in plasma. NeuroRx 1, 226-234.
- Jennum P, K. J. (July 2011). Health, social and economical consequences of sleep-disordered breathing: a controlled national study. . *Thorax*, 66(7):560-6.
- Jha A, W. A.-F. (Jan-Feb 2008). A randomized trial of modafinil for the treatment of fatigue and excessive daytime sleepiness in individuals with chronic traumatic brain injury. . *J Head Trauma Rehabil*, 23 (1):52-63.
- JJ, G. (August 2008). Treatment of circadian rhythm sleep disorders with light. *Ann Acad Med Singapore*, 37(8):669-76.
- Kalmar K, N. T.-R. (2008). Feasibility and utility of a brief neuropsychological test battery for use during acute inpatient rehabilitation after TBI. *Arch Phys Med Rehabil*, 89:94.
- Kayihan, G. C. (2010). Gulf War agents trigger discrete transcriptional changes in human neuronal cells. *Toxicological & Environmental Chemistry*, 92, 1783-1799.
- Krueger, F. P. (2011). The role of the Met66 brain-derived neurotrophic factor allele in the recovery of executive functioning after combat-related traumatic brain injury. *J Neurosci*, 31, 598-606.
- Lakhan, S. E. (2009). Schizophrenia genomics and proteomics: are we any closer to biomarker discovery? . *Behav Brain Funct*, 5, 2.
- Lakshmanan, R. L. (2010). Metabolic crisis after traumatic brain injury is associated with a novel microdialysis proteome. . *Neurocrit Care*, 12, 324-336.
- Larson EB, Z. F. (2010). The effect of sleep medications on cognitive recovery from traumatic brain injury. *J Head Trauma Rehabil*, 25(1):61-7.
- Lim J, D. D. (2008). Sleep deprivation and vigilant attention. Ann N Y Acad Sci, 1129:305-22.
- Lista, S. F. (2013). Blood and plasma-based proteomic biomarker research in Alzheimer's disease. *Prog Neurobiol*, 101-102, 1-17.
- Lockley SW, G. J. (2006). Circadian photoreception: Spotlight on the brain. Curr Biol, 16(18):R795-7.
- Longordo F, K. C. (2009). Consequences of sleep deprivation on neurotransmitter receptor expression and function. *European Journal of Neuroscience*, 29:1810-9.
- Luis, C. A. (2009). Serum beta-amyloid correlates with neuropsychological impairment. *Neuropsychol Dev Cogn B Aging Neuropsychol Cogn*, 16, 203-218.
- Luis, C. A.-G. (2011). Feasibility of Predicting MCI/AD Using Neuropsychological Tests and Serum β-Amyloid. *Int J Alzheimers Dis*.
- Makley MJ, E. J. (2008). Prevalence of sleep disturbance in closed head injury patients in a rehabilitation uni. *Neurorehabil Neural Repair.*, 341-7.
- Makley MJ, J.-G. L. (2009). Return of memory and sleep efficiency following moderate to severe closed head injury. *Neurorehabil Neural Repair*, 23 (4):320-6.

- Marshall L, H. H. (2006). Boosting slow oscillations during sleep potentiates memory. *Nature*, 444:610-613.
- Martins-de-Souza, D. M. (2010). Proteome analysis of the thalamus and cerebrospinal fluid reveals glycolysis dysfunction and potential biomarkers candidates for schizophrenia. *J Psychiatr Res*, 44, 1176-1189.
- Mathias JL, A. P. (2012;13). Prevalence of sleep disturbances, disorders, and problems following traumatic brain injury: A meta analysis. . *Sleep Med*, 898-905.
- McDermott CM, L. G. (2003). Sleep deprivation causes behavioral, synaptic, and membrane excitability alterations in hippocampual neurons. *J. Neuroscience*, 23:9687-95.
- Melyan Z, T. E. (2005). Addition of human melanopsin renders mammalian cells photoresponsive. *Nature*, 433(7027):741-745.
- Mishima K, O. M. (1994). Morning bright light therapy for sleep and behavior disorders in elderly patients with dementia. *Acta Psychiatr Scand*, 89(1):1-7.
- Morgenthaler TI, L.-C. T. (2007, Nov 30). An American Academy of Sleep Medicine Report: Practice parameters for the clinical evaluation and treatment of circadian rhythm sleep disorders. *Sleep*, 30(11), 1445-59.
- Nakase-Richardson R, K. T. (2012). The role of sleep in maximizing rehabilitation outcome: Experience of three VHA programs. Recorded symposium. 2012 American Psychological Association Annual Conference.
- Nakase-Richardson R, S. D. ( (under review)). Does White Light Exposure Differ Among Acute Neurorehabilitation Admissions?
- Nakase-Richardson R, S. D. ((Under Review)). Feasibility of Polysomnography Objective Sleep Assessment in the Acute Moderate to Severe Traumatic Brain Injury Patient.
- Nakase-Richardson R, S. M. (2013). Prospective evaluation of the nature, course, and impact of acute sleep abnormality following TBI. *Archives of Physical Medicine and Rehabilitation*, 875-82.
- Nakase-Richardson R, S. M. (2013). Prospective evaluation of the nature, course, and impact of acute sleep abnormality following TBI . *Archives of Physical Medicine and Rehabilitation 2013;*, 94 (5): 875-82.
- National Data and Statistical Center. (2013, August 1). *VA Polytrauma Center Database Syllabus*. Retrieved from Traumatic Brain Injury Model Systems National Database: www.tbindscva.org/Syllabus.aspx
- Neikrug AB, R. M.-I. (2012). Bright light therapy protects women from circadian rhythm desynchronization during chemotherapy for breast cancer. *Behav Sleep Med*, 10(3):202-16.
- Netzer NC, S. R. (1999). Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome. *Ann Intern Med*, 485-491.
- Ohayon MM, R. C. (2009). 3rd. Epidemiological and clinical relevance of insomnia diagnosis algorithms according to the DSM-IV and the International Classification of Sleep Disorders (ICSD). *Sleep Med.*, 952-60.
- Okonkwo, D. O. (2013). GFAP-BDP as an Acute Diagnostic Marker in Traumatic Brain Injury: Results from the prospective TRACK-TBI Study. *J Neurotrauma*.
- Orff HG, A. L. (2009). Traumatic brain injury and sleep disturbance: a review of current research. *J Head Trauma Rehabilitation*, 155-65.
- Ouellet MC, M. C. (2007). Efficacy of cognitive-behavioral therapy for insomnia associated with traumatic brain injury: a single-case experimental design. *Arch Phys Med Rehabil*, 1581-92.
- Ouellet MC, S. J. (2004). Insomnia following traumatic brain injury: a review. *Neurorehabilitation Neural Repair*, 18 (4): 187-98.
- Pineda, J. L. (2007). Clinical significance of alphaII-spectrin breakdown products in cerebrospinal fluid after severe traumatic brain injury. *J Neurotrauma*, 24, 354-366.
- Ponsford JL, Z. P.-N. (May-Jun 2012). Fatigue and sleep disturbance following traumatic brain injury--their nature, causes, and potential treatments. *J Head Trauma Rehabil*, 27(3):224-33.
- R., N.-R. (2012). Sleep disturbance during acute inpatient rehabilitation. *Recorded symposium: Wrestling with Hypnos: Sleep, Wake, and Fatigue After TBI.* 2012 American Congress of Rehabilitation Medicine Annual Conference.

- RD., L. (Jan 2005). What is the optimal implementation of bright light therapy for seasonal affective disorder (SAD)? *J Psychiatry Neurosci*, 30(1):72.
- Reeves GM, N. G. (2012). Improvement in depression scores after 1 hour of light therapy treatment in patients with seasonal affective disorder. *J Nerv Ment Dis.*, 51-55.
- Revell VL, B. H. (Jan 2006). Advancing human circadian rhythms with afternoon melatonin and morning intermittent bright light. *J Clin Endocrinol Met*, 91(1):54-9.
- Riemersma-van der Lek RF, S. D. (2008). Effect of bright light and melatonin on cognitive and noncognitive function in elderly residents of group care facilities: a randomized controlled trial. *JAMA*, 2642-55.
- Roses, A. &. (1997). ApoE, Alzheimer's disease, and recovery from brain stress. *Ann N Y Acad Sci*, 826, 200-212.
- Schneider Soares, F. M. (2012). Interleukin-10 is an independent biomarker of severe traumatic brain injury prognosis. *Neuroimmunomodulation*, 19, 377-385.
- Services, S. A. (1982). Symbol digit modalities test: Manual. Los Angeles: Western Psychological.
- Sheinerman, K. S. (2012). Plasma microRNA biomarkers for detection of mild cognitive impairment. *Aging*, 4, 590-605.
- Sherer M, Y. S.-R. (2009). Patterns of recovery of posttraumatic confusional state in neurorehabilitataion admissions after traumatic brain injury. *Arch Phys Med Rehabil*, 90(10):1749-54.
- Shum D, M. K. (1990). Construct validity of eight tests of attention: Comparison of normal and closed head injured samples. *Clinical Neuropsychologist*, 4(2):151-62.
- Silva, M., Nakase-Richardson, R., M, S., SD, B., CC, E., & SA, Y. (2012). Posttraumatic confusion predicts patient cooperation during traumatic brain injury rehabilitation. *Am J Phys Med Rehabil*, 91 (10):890-3.
- Sjösten N, K. M. (July 2009). Obstructive sleep apnoea syndrome as a predictor of work disability. *Respir Med*, 103(7):1047-55.
- Smith MR, R. V. (Mar 2009). Phase advancing the human circadian clock with blue-enriched polychromatic light. *Sleep Med*, 10(3):287-94.
- State University of New York at Buffalo. (1997). Guide for the Uniform Data Set for Medical Rehabilitation (including the FIM(TM) instrument. Buffalo, NY, United States.
- Terman M, T. J. (2005). Light therapy for seasonal and nonseasonal depression: efficacy, protocol, safety, and side effects. *CNS Spectr*, 10(8):647-63.
- Traumatic Brain Injury Model Systems. (2013, August 1). *Identification of Subjects*. Retrieved from National Data and Statistical Center: www.tbindsc.org/SOP.aspx
- Trzepacz PT, M. D. (2001). Validation of the Delirium Rating Scale Revised: Comparison with the Delirium Rating Scale and the Cognitive Test for Delirium. *J Neuropsychiatr Clin Neuroscience*, 13:229-42.
- Turner PL, M. M. (2008). Circadian photoreception: Ageing and the eye's important role in systemic health. *Br J Ophthalmol*, 92(11):1439-1444.
- Verma A, A. V. (2007). Sleep disorders in chronic traumatic brain injury. J Clin Sleep Med, 3(4):357-62.
- Viant, M. R. (2005). An NMR metabolomic investigation of early metabolic disturbances following traumatic brain injury in a mammalian model. *NMR Biomed*, 18, 507-516.
- Walder, B. R. (2013). The prognostic significance of the serum biomarker H-FABP in comparison with S100b in severe traumatic brain injury. *J Neurotrauma*.
- Wäljas M, I. G. (2012). Reliability, validity and clinical usefulness of the BNI fatigue scale in mild traumatic brain injury. *Brain Inj*, 26:972-8.
- Walker, M. (2009). The role of sleep in cognition and emotion. Ann New York Acad Science, 1156:168-97.
- Waters, R. &. (2005). Genetic influences on outcome following acute neurological insults. . *Curr Opin Crit Care*, 11, 105-110.
- Watson NF, D. S. (2007). Hypersomnia following traumatic brain injury. J Clin Sleep Med, 3(4):363-8.
- Watson, D. L. (1988). Development and validation of brief measures of positive and negative affect: The PANAS scales. *Journal of Personality and Social Psychology*, 54 (6), 1063-1070.

- Webster JB, B. K. (March 2001). Sleep apnea in adults with traumatic brain injury: a preliminary investigation. *Arch Phys Med Rehabilitation*, 316-21.
- Whitmore RG, T. J. (2012). Is aggressive treatment of traumatic brain injury cost-effective? . *J Neurosurg* , 116(5):1106-13.
- Wilde MC, C. R. (2007). Cognitive impairment in patients with traumatic brain injury and obstructive sleep apnea. *Arch Phys Med Rehabil*, 88: 1284-8.
- Wirz-Justice A, T. M. (2012). Chronotherapeutics (light and wake therapy) as a class of interventions for affective disorders. *Handb Clin Neurol*, 697-713.
- Wood RL, M. J. (1999). Clinical and cost effectiveness of postacute neurobehavioural rehabilitation. *Brain Inj*, 13(2):69-88.
- Yordoova J, K. V. (2012). Increased alpha (8-12 Hz) activity during slow wave sleep as a marker for the transition from implicit knowledge to explicit insight. *J Cogn Neurosci*, 24:119-32.
- Zeitzer JM, D. D. (2000). Sensitivity of the human circadian pacemaker to nocturnal light: melatonin phase resetting and suppression. *J Physiol*, 526 Pt 3:695-702.
- Zhao, W. H. (2013). Decreased level of olfactory receptors in blood cells following traumatic brain injury and potential association with tauopathy. *J Alzheimers Dis*, 34, 417-429.
- Zhou W, X. D. (Apr 25 2008). Meta-analysis of APOE4 allele and outcome after traumatic brain injury. *J Neurotrauma*, (4):279-90.
- Zollman FS, C. C. (2010). Actigraphy for assessment of sleep in traumatic brain injury: case series, review of the literature and proposed criteria for use. *Brain Inj*, 24 (5):748-54.
- Zollman FS, L. E.-T. (Mar-Apr 2012). Acupuncture for treatment of insomnia in patients with traumatic brain injury: a pilot intervention study. *J Head Trauma Rehabi*, 27(2):135-42.
- Zunzunegui C, G. B. (2011). Sleep disturbance impairs stroke recovery in the rat. . Sleep, 34(9):1261-9.

## **Appendix**

- Inclusion/Exclusion Checklist
- Makley Sleep Scale Form
- Berlin Questionnaire
- Del-R-98, Question 1 Form
- Functional Independence Measure (FIM)<sup>TM</sup>
- PANAS
- Karolinska Sleepiness Scale
- Barrow Neurological Institute Fatigue Scale
- Quarterly Staff Survey (a.k.a. Clinician Feasibility Survey)
- Overview of Study Figure

#### **TWILIGHT Study Inclusion and Exclusion Checklist**

## **Inclusion Criteria** Must meet all of the criteria below ☐ Have experienced a moderate to severe TBI. Defined by any of the following: 1) Loss of Consciousness greater than 30 minutes. 2) Emergency Room admission with a Glasgow Coma Scale of 12 or below. 3) Intracranial abnormalities on imaging. 4) Post-traumatic amnesia that lasts more than 24 hours. ☐ Admitted to acute inpatient rehabilitation unit at Harborview Medical Center within 3 months of their Traumatic Brain Injury. ☐ Able to communicate in English. ☐ Between the ages of 18 and 70 years old **Exclusion Criteria** Unable to enroll if any of the following are true ☐ Complete blindness ☐ Absence of eye opening or disorders of consciousness (Rancho level 1-3) Does not have sleep disturbance (rating of "0" on item one of the *DelRS-R98*. If has a rating of "0", but if taking sleep medication in the last 72 hours, then include) ☐ Tetraplegia with less than antigravity strength in all myotomes caudal to C6 level given the limitations on measuring movements with actigraphy in this population (i.e. cannot reliably detect upper extremity or lower extremity movement with this level of paralysis). ☐ Past medical history of retinal pathology ☐ Past medical history of light sensitivity ☐ Past medical history of narcolepsy ☐ Past medical history of bipolar disorder ☐ Past medical history of obstructive sleep apnea ☐ Suspected sleep apnea. (Determined by administering the Berlin questionnaire) ☐ Current medical orders indicated for night time sleep disruption (e.g. chest PT, MIE q2 hours of meds that disrupt sleep)". For these subjects, may re-approached if the medical orders are no longer in place.

## TWILIGHT STUDY

| ☐ Was watch verified as on? | Staff Initials | Date: |
|---|---|---|
| | Makley Sleep Scale Form<br>Clinician rating | |

| | | | imician raung | | |
|---|---|---|---|---|---|
| Time | Rounding | Sleep Rat | ing Given Observa | tion in the Last Ho | our |
| | Initials | (circle) | | | |
| 2200 | | 0 | 1 | 2 | 3 |
| 2300 | | 0 | 1 | 2 | 3 |
| 0000 | | 0 | 1 | 2 | 3 |
| 0100 | | 0 | 1 | 2 | 3 |
| 0200 | | 0 | 1 | 2 | 3 |
| 0300 | | 0 | 1 | 2 | 3 |
| 0400 | | 0 | 1 | 2 | 3 |
| 0500 | | 0 | 1 | 2 | 3 |
| 0600 | | 0 | 1 | 2 | 3 |
| Ratings: | | Asleep | Drowsy/falling<br>asleep | Drowsy/waking<br>up | awake |

| Where there any adverse events or effects? $\square \text{Yes } \square \text{No}$ | Source: |
|---|---|
| If yes, please explain | |

## Makley Sleep Log guidelines and FAQ's

#### **Data collection**

- 1. The sleep log can by collected by nurses or MA staff
- 2. Clinical staff will do data collection rounding on an hourly basis and rate the patient accordingly with a 0,1,2 or 3
- 3. The rating for each hour is the clinical staffs best assessment of observed sleep/non-sleep state based on how they were found, not what was being done clinically, if anything
- 4. Hourly ratings may be collected on paper or electronically
- 5. Sleep log for the first night, along with any and all information about the participant's sleep over the last 3 nights will be used to randomize. Information about the participant's sleep will be asked of any family or friends' present, clinical staff, medical chart review, and nursing notes. Please look to see if the participant has or is on any sleep medications in the past 72 hours.
- 6. Once the research staff has all information, they will rate the participant using the DelRS-98 item #1 to score their severity of sleep
- 7. Data may need to be used to reconcile actigraphy data if there are questions
- 8. Research staff should collect the sleep logs on a daily basis and place a copy in the participants file (deidentified)

## FAQ's

- 1. Clinically what's the difference between 1 (falling asleep) and 2 (waking up) in the setting of night time rounds? Can we tell? **Answer**: Make your best clinically assessment. If patient is fully asleep then score = 0, if patient is fully awake then score = 3.
- 2. What do we do with missing hours on a sleep log? **Answer**: note it as missing data; follow-up with staff training/study education.
- 3. What do we do when a sleep log is entirely missing? **Answer**: keep looking to see if it can be found; include notation in case notes; follow-up with staff training/study education.
- 4. Staff says a patient slept fine but family notes the patient was restless overnight, what data do we take for rating of sleep disturbance in the study? **Answer**: Clinically we know that patients/subjects will be observed at different time points and that the type and quality of observations will be variable. Research staff should collect all available data and make their best summary of presence/absence of ANY sleep changes and if present the rating of severity (using the Del-RS-R 98 item 1) considering that this type of data is generally additive to describe what's happened overnight and not necessarily either/or. To score a subject as having no sleep disturbance there should be no clinical data that says the patient didn't sleep perfectly well (i.e. patient/caregiver/family report is all that sleep was fine, no medications given).

35

Manual of Procedures: TWILIGHT Study Rev: 9/2/2014

| _ | ESTIONNAIRE | <b>A</b> | M-1- / F1- | |
|---|---|---|---|---|
| | Weight (kg) | | _ Male / Female | |
| Please choose | the correct response to each | question. | | |
| CATEGORY | 1 | | | |
| 1. Do you sno | re? | | | |
| · | a. Yes | b. <b>1</b> | No | c. Don't know |
| | If you snore: | | | |
| | 2. Your snoring is: | | | |
| | a. Slightly louder than b | reathing | | |
| | b. As loud as talking | | | |
| | c. Louder than talking | | | |
| | d.Very loud – can be he | eard in adjacen | nt rooms | |
| 3. How often | do you snore | | | |
| | Nearly every day | | | |
| b. | 3-4 times a week | | | |
| c. | 1-2 times a week | | | |
| d. | 1-2 times a month | | | |
| e. | Never or nearly never | | | |
| 4 ** | | 1.0 | | |
| • | noring ever bothered other | r people? | | |
| | Yes | | | |
| | No<br>Day't Know | | | |
| С. | Don't Know | | | |
| 5. Has anyone | e noticed that you quit brea | athing durin | g your sleep? | |
| | Nearly every day | O | <b>1</b> | |
| b. | 3-4 times a week | | | |
| c. | 1-2 times a week | | | |
| d. | 1-2 times a month | | | |
| e. | Never or nearly never | | | |
| CATECODY | <b>.</b> . | | | |
| CATEGORY | do you feel tired or fatigue | d ofter your | sloop? | |
| | Nearly every day | u aitei youi | sieep. | |
| | 3-4 times a week | | | |
| | 1-2 times a week | | | |
| | 1-2 times a week | | | |
| | Never or nearly never | | | |
| e. | Never of flearly flever | | | |
| 7. During you | ır waking time, do you feel | tired, fatigu | ed or not up to par? | |
| a. | Nearly every day | | _ | |
| b. | 3-4 times a week | | | |
| c. | 1-2 times a week | | | |
| d. | 1-2 times a month | | | |
| e. | Never or nearly never | | | |

 $8. \ Have \ you \ ever \ nodded \ off \ or \ fallen \ as leep \ while \ driving \ a \ vehicle?$ 

- a. Yes
- b. No

## *If yes:*

## 9. How often does this occur?

- a. Nearly every day
- b. 3-4 times a week
- c. 1-2 times a week
- d. 1-2 times a month
- e. Never or nearly never

## **CATEGORY 3**

## 10. Do you have high blood pressure?

- a. Yes
- b. No
- c. Don't know

#### Rating Sleep-Wake cycle disturbance:

Question 1 is utilized in this study

#### DELIRIUM RATING SCALE-R-98 (DRS-R-98)

This is a revision of the Delirium Rating Scale (Trzepacz et al. 1988). It is used for initial assessment and repeated measurements of delirium symptom severity. The sum of the 13 item scores provides a severity score. All available sources of information are used to rate the items (nurses, family, chart) in addition to examination of the patient. For serial repeated ratings of delirium severity, reasonable time frames should be chosen between ratings to document meaningful changes because delirium symptom severity can fluctuate without interventions.

#### **DRS-R-98 SEVERITY SCALE**

#### 1. Sleep-wake cycle disturbance

Rate sleep-wake pattern using all sources of information, including from family, caregivers, nurses' reports, and patient. Try to distinguish sleep from resting with eyes closed.

- Not present
- 1. Mild sleep continuity disturbance at night or occasional drowsiness during the day
- Moderate disorganization of sleep-wake cycle (e.g., falling asleep during conversations, napping during the day or several brief awakenings during the night with confusion/behavioral changes or very little nighttime sleep)
- Severe disruption of sleep-wake cycle (e.g., day-night reversal of sleep-wake cycle or severe circadian fragmentation with multiple periods of sleep and wakefulness or severe sleeplessness.)

#### 2. Perceptual disturbances and hallucinations

Illusions and hallucinations can be of any sensory modality. Misperceptions are "simple" if they are uncomplicated, such as a sound, noise, color, spot, or flashes and "complex" if they are multidimensional, such as voices, music, people, animals, or scenes. Rate if reported by patient or caregiver, or inferred by observation.

- 0. Not present
- Mild perceptual disturbances (e.g., feelings of derealization or depersonalization; or patient may not be able to discriminate dreams from reality)
- Illusions present
- 3. Hallucinations present

#### 3. Delusions

Delusions can be of any type, but are most often persecutory. Rate if reported by patient, family or caregiver. Rate as delusional if ideas are unlikely to be true yet are believed by the patient who cannot be dissuaded by logic. Delusional ideas cannot be explained otherwise by the patient's usual cultural or religious background.

- 0. Not present
- 1. Mildly suspicious, hypervigilant, or preoccupied
- 2. Unusual or overvalued ideation that does not reach delusional proportions or could be plausible
- 3. Delusional

#### 4. Lability of affect

Rate the patient's affect as the outward presentation of emotions and not as a description of what the patient feels.

- Not present
- 1. Affect somewhat altered or incongruent to situation; changes over the course of hours; emotions are mostly under self-control
- Affect is often inappropriate to the situation and intermittently changes over the course of minutes; emotions are not consistently under self-control, though they respond to redirection by others
- Severe and consistent disinhibition of emotions; affect changes rapidly, is inappropriate to context, and does not respond to redirection by others

#### 5. Language

Rate abnormalities of spoken, written or sign language that cannot be otherwise attributed to dialect or stuttering. Assess fluency, grammar, comprehension, semantic content and naming. Test comprehension and naming nonverbally if necessary by having patient follow commands or point.

- 0. Normal language
- 1. Mild impairment including word-finding difficulty or problems with naming or fluency
- 2. Moderate impairment including comprehension difficulties or deficits in meaningful communication (semantic content)
- 3. Severe impairment including nonsensical semantic content, word salad, muteness, or severely reduced comprehension

FIM-**Functional** Independence Measure SELF CARE ITEMS: ADMISSION DISCHARGE 7=Complete Independence (Timely, safely) 1. Feeding 2. Grooming ..... 6=Modified Independence (Extra time, device) 5=Supervision (pt does 100%) 3. Bathing 4. Dressing Upper Body ..... 4=Minimal Assistance (pt >75% of task) 5. Dressing Lower Body ..... 3=Moderate Assistance (pt 50-74% of task) 6. Toileting 2=Maximum Assistance (pt 25-49% of task) 1=Total Assistance (pt<25% of task) SPHINCTER CONTROL: 0=Activity does not occur. (Use only at admission and only for #1-6,10-15; else use code "9".) 8. Bladder Management ..... a. Level of assistance...... 8=N/A, pt walking/not using wheelchair. b. Frequency of accidents..... (only for item #14b) Bowel Management ...... 9=Unknown / assessed at >72 hours / activity does a. Level of assistance..... not occur (see instructions in code "0", above). b. Frequency of accidents 66=Data not available with new (1/1/02) scoring. (Use only at admission and only for #1-8a, 9, 9a, MOBILITY ITEMS: 10-15) Transfer Technique 10. Bed. Chair. Wheelchair ..... Use with 8b and 9b 11. Toilet 7=No accidents 12. Tub or Shower ..... 6=No accidents; uses device (catheter, ostomy) 5=One accident in the past 7 days 4=Two accidents in the past 7 days Locomotion 14a. Walking on admission 3=Three accidents in the past 7 days 14b. Wheelchair on admission ..... 2=Four accidents in the past 7 days 14. Walking/Wheelchair-discharge (w/c/9) ..... 1=Five or more accidents in the past 7 days 15. Stairs ..... 9= Unknown / assessed at >72 hours 66=Variable did not exist COMMUNICATIONS: Comprehension ...(a/v/b/9) ........ 18. Expression ..... (v/n/b/9) ....... PSYCHOSOCIAL ADJUSTMENT ITEMS: 22. Social Interaction .....

39

COGNITIVE FUNCTION:

#### PANAS Questionnaire

This scale consists of a number of words that describe different feelings and emotions. Read each item and then list the number from the scale below next to each word. Indicate to what extent you feel this way right now, that is, at the present moment *OR* indicate the extent you have felt this way over the past week (circle the instructions you followed when taking this measure)

| 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|
| Very Slightly or Not<br>at All | A Little | Moderately | Quite a Bit | Extremely |

| 1. Interested | 11. Irritable |
|-----------------|----------------|
| 2. Distressed | 12. Alert |
| 3. Excited | 13. Ashamed |
| 4. Upset | 14. Inspired |
| 5. Strong | 15. Nervous |
| 6. Guilty | 16. Determined |
| 7. Scared | 17. Attentive |
| 8. Hostile | 18. Jittery |
| 9. Enthusiastic | 19. Active |
| 10. Proud | 20. Afraid |

#### Scoring Instructions:

Positive Affect Score: Add the scores on items 1, 3, 5, 9, 10, 12, 14, 16, 17, and 19. Scores can range from 10 - 50, with higher scores representing higher levels of positive affect. Mean Scores: Momentary = 29.7 (SD = 7.9); Weekly = 33.3 (SD = 7.2)

Negative Affect Score: Add the scores on items 2, 4, 6, 7, 8, 11, 13, 15, 18, and 20. Scores can range from 10 - 50, with lower scores representing lower levels of negative affect. Mean Score: Momentary = 14.8 (SD = 5.4); Weekly = 17.4 (SD = 6.2)

Copyright © 1988 by the American Psychological Association. Reproduced with permission. The official citation that should be used in referencing this material is Watson, D., Clark, L. A., & Tellegan, A. (1988). Development and validation of brief measures of positive and negative affect: The PANAS scales. Journal of Personality and Social Psychology, 54(6), 1063–1070.

| BASELINE | Pt. not able to report $\Box$ |
|----------|-------------------------------|
|----------|-------------------------------|

## Sleepiness Scale: (Karolinska Sleepiness Scale)

Here are some descriptors about how alert or sleepy you might be feeling right now. Which one corresponds to the statement describing how you feel at this moment?

- i. Extremely alert
- ii. Very alert
- iii. Alert
- iv. Rather Alert
- v. Neither alert nor sleepy
- vi. Some signs of sleepiness
- vii. Sleepy, but no difficulty remaining awake
- viii. Sleepy, some effort to keep alert

| Pre Light Treatment |
|---------------------|
|---------------------|

| Date: | Score: |
|-------|--------|

## **BASELINE**

## **Barrow Neurological Institute Fatigue Scale**

Pt. not able to report  $\Box$ 

Please rate the extent to which each of the items below has been a problem for you since your injury. You should choose only ONE number from 0-7 on the scale below when making your response.

| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
|---|---|---|---|---|---|---|---|
| Rarely a problem | | Occasional problem but not frequent | | quent<br>olem | A pi | roblem most<br>the time | of |

- 1. How difficult is it for me to maintain my energy throughout the day?
- 2. How difficult is it for me to participate in activities because of fatigue?
- 3. How difficult is it for me to stay awake during the day?
- 4. How difficult is it for me to complete a task without becoming tired?
- 5. How difficult is it for me to stay alert during activities?
- 6. How difficult is it for me to build my energy level once I wake up in the morning?
- 7. How difficult is it for me to stay out of my bed during the day?
- 8. How difficult is it for me to stay alert when I am not involved in something?
- 9. How difficult is it for me to attend to something without becoming sleepy?
- 10. How difficult is it for me to last the day without taking a nap?

## 11. Please circle your OVERALL level of fatigue since your injury:

| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
|---------|---|---|---|---|---|---|---|---|---|---------|
| No | | | | | | | | | | Severe |
| problem | | | | | | | | | | Problem |



## **Quarterly Staff Survey**

If you have been involved in the care of a patient enrolled in the TWILIGHT Study in the past three months please answer the questions below.

| Date: | | | | |
|---|---|---|---|---|
| Please check one: | | | | |
| ☐ Rehabilitation Nu | rse | | | |
| ☐ Rehabilitation The | erapist (PT, OT, SLP, T | R) | | |
| □ Other | | | | |
| Please indicate whether y | ou agree or disagree | with the following statement | s: | |
| Q1: It was easy to integra | ate light therapy into | patient care. | | |
| 1 | 2 | 3 | 4 | 5 |
| Strongly Disagree | Disagree | Neither agree or disagree | Agree | Strongly Agree |
| Q2: Light therapy did not increase my work load. | | | | |
| 1 | 2 | 3 | 4 | 5 |
| Strongly Disagree | Disagree | Neither agree or disagree | Agree | Strongly Agree |
| · | | • | | |

Q3: Light therapy should be offered as a routine treatment option in in-patient rehabilitation.

| 1 | 2 | 3 | 4 | 5 |
|-------------------|----------|------------------|-------|----------------|
| Strongly Disagree | Disagree | Neither agree or | Agree | Strongly Agree |
| | | disagree | | |

**Comments?** 

## **Overview for Study Participants**

